

### Statistical Analysis Plan

NCT Number: NCT05543187

Title: An Open-Label, Phase 3 Study to Evaluate the Efficacy and Safety of TAK-625 in

the Treatment of Subjects With Progressive Familial Intrahepatic Cholestasis

Study Number: TAK-625-3002

Document Version and Date: Version 1.0 / 5-Sep-2025

Certain information within this document has been redacted (ie, specific content is masked irreversibly from view) to protect either personally identifiable information or company confidential information.



## STATISTICAL ANALYSIS PLAN for Final Analysis

Study Number: TAK-625-3002

aute the Effica
sive Familial Intra.

Phase: 3
Version: 1.0
Date: 5-Sep-2025

ased on:

Protocol Version: Amendment 2
Protocol Date: 08-Dec-2022 Study Title: An Open-Label, Phase 3 Study to Evaluate the Efficacy and Safety of TAK-625 in the Treatment of Subjects with Progressive Familial Intrahepatic Cholestasis

Prepared by:

Based on:

98. For non

### CONFIDENTIAL PROPERTY OF TAKEDA

This document is a confidential communication of Takeda. Acceptance of this document constitutes the agreement by the recipient that no information contained herein will be published or disclosed without written authorization from Takeda.

### **REVISION HISTORY**

| [Original version] [Not Applicable] |
|---|
| and subject to the applicable to |
| REVISION HISTORY Version Approval Date Primary Rationale for Revision [Original version] [Not Applicable] Not Applicable Applicable Primary Rationale for Revision [Original version] [Not Applicable] |

### **TABLE OF CONTENTS**

| 1.0 | OBJE | CTIVES, ENDPOINTS AND ESTIMANDS | 8 |
|---|---|---|---|
| 1. | | jectives | |
| | 1.1.1 | Primary Objective | 20, |
| | 1.1.2 | Primary Objective | (S) |
| | 1.1.3 | Additional Objective(s) | |
| 1.3 | 2 En | dpoints | , 2 <sup>(2)</sup> |
| | 1.2.1 | Additional Objective(s) dpoints Primary Endpoint(s) Secondary Endpoint(s) .2.1 Key Secondary Endpoints(s) | ,<br>8 |
| | 1.2.2 | Secondary Endpoint(s) | 8 |
| | 1.2 | .2.1 Key Secondary Endpoints(s) | 8 |
| | 1.2 | .2.2 Secondary Endpoint(s) | 8 |
| | | × | |
| | 1.2.4 | Safety Endpoints | |
| | 1.2.5 | Other Endpoints | 10 |
| | 1.2 | Safety Endpoints Other Endpoints .5.1 PK Endpoint timand(s) Y DESIGN | 10 |
| 1 | 3 Est | timand(s) | 10 |
| 2.0 | STUD | Y DESIGN | 10 |
| 3.0 | STAT | STICAL HYPOTHESES AND DECISION RULES | 12 |
| 4.0 | SAMP | LE-SIZE DETERMINATION | 12 |
| 5.0 | ANAL | YSIS SETS | 12 |
| 5. | 1 All | Subjects Who Signed the Informed Consent Form | 12 |
| 5.2 | 2 All | Subjects Who Did Not Enter the Treatment Period | 12 |
| 5 | 3 Sat | fety Analysis, Set | 13 |
| 5.4 | 4 Int | ention-to-treat set (ITT) | 13 |
| 5 | 5 Pei | r-Protocol Analysis Set (PPS) | 13 |
| 6.0 | STAT | ISTICAL ANALYSIS | 13 |
| 6. | 1 Ge | neral Considerations | 13 |
| 6.2 | 2 An | alysis Approach | 15 |
| C | 6.2.1 | Analysis Cohort | |
| (0) | 6.2.2 | Analysis Approach for Continuous Efficacy Endpoints | 15 |
| C | 6.2.3 | Analysis Approach for Binary Efficacy Endpoints | 15 |
| • | 6.2.4 | Analysis Approach for Time-to-Event Efficacy Endpoints | 15 |
| 6 | 3 Dis | sposition of Subjects | 16 |
| | 6.3.1 | Study Information | 16 |
| | 632 | Disposition of Subjects | 16 |

| | (22 | D ( 1D 1) 1 1 1 1 C ( | 1.7 |
|---|---|---|---|
| | 6.3.3 | Protocol Deviations and Analysis Sets | |
| | 6.3. | - 6 | |
| | 6.3. | 3.2 Analysis Sets | 17 |
| 6. | 4 Cor | ent of Exposure and Compliance | 8 |
| 6. | 5 Ext | ent of Exposure and Compliance | |
| 6. | 6 Effi | cacy Analysis | 29 |
| | | <b>√</b> . | |
| 6. | 7 Safe | ety Analysis | 22 |
| | 6.7.1 | | |
| | 6.7. | 1.1 Overview of Treatment-Emergent Adverse Events | 22 |
| | 6.7. | | |
| | 6.7.2 | Clinical Laboratory Evaluations | |
| | 6.7. | 2.1 Laboratory Tests other than Urinalysis | 25 |
| | 6.7. | 2.2 Urinalysis | 25 |
| | 6.7.3 | Vital Signs, Weight and Height | 26 |
| | 6.7.4 | ECGs | 27 |
| | 6.7.5 | Displays of Treatment-Emergent Adverse Events (Japanese) | 27 |
| 6. | 8 Pha | rmacokinetic, Pharmacodynamic, and Biomarker Analyses | 28 |
| | 6.8.1 | Pharmacokinetic Analysis | 28 |
| 6. | 9 Oth | er Analyses | 28 |
| | 6.9.1 | Analyses for Overall Supplemental Cohort | |
| | 6.9.2 | Analyses for All Cohorts Combined | |
| 7.0 | REFER | BNCES | |
| 8.0 | CHAN | GES TO PROTOCOL PLANNED ANALYSES | 28 |
| 9.0 | APPEN | | |
| 9. | 1 Cha | inges From the Previous Version of the SAP | |
| 9. | | a Handling Conventions | |
| $k_{\mathbf{X}}$ | 9.2.1 | Definition of Study Days | |
| | 9.2.2 | Definition of Study Visit Windows | |
| | 9.2. | • | |
| | 9.2. | | |
| | 9.2. | 1 | |
| | | C) | |

### ABBREVIATIONS

ΑE adverse event

**AECI** adverse event of clinical interest

AFP alpha-fetoprotein **ALP** alkaline phosphatase ALT alanine aminotransferase ANCOVA analysis of covariance APRI AST to platelet ratio index

aPTT activated partial thromboplastin time

AST aspartate aminotransferase 7αC4 7α-hydroxy-4-cholesten-3-one

BMI body mass index **BUN** blood urea nitrogen CBC complete blood count CI confidence interval

**ECG** Electrocardiogram

fibroblast growth factor 190 FGF-19

fibrosis-4 FIB-4

gamma-glutamyl transferase **GGT** hepatocellular carcinoma **HCC** 

high density lipoprotein-cholesterol HDL-C

health-related quality of life **HRQoL** 

ItchRO Observer ItchRO(Obs) ItchRO Patient ItchRO(Pt) ITT intention-to-treat set

**KM** Kaplan-Meier

low density lipoprotein-cholesterol

lower limit of normal

last observation carried forward

LSV least square means lipid soluble vitamin

**MCH** mean corpuscular hemoglobin

**MCHC** mean corpuscular hemoglobin concentration

**MCV** mean corpuscular volume MedDRA Medical Dictionary for Regulatory Activities

**MITT** modified intention-to-treat set **PEBD** partial external biliary diversion

**PFIC** progressive familial intrahepatic cholestasis

PK pharmacokinetic

**PPS** per-protocol analysis set PRO patient-reported outcomes

PT preferred term 25th percentile Q1 Q3 75th percentile

QT interval corrected using Bazett's formula QTcB QT interval corrected using Fridericia's formula QTcF only and sul

QOL quality-of-life

retinol binding protein RBP SAE serious adverse event SAP statistical analysis plan

sBAserum bile acid

**SGOT** serum glutamic-oxaloacetic transaminase serum glutamic-pyruvic transaminase **SGPT** 

SOC system organ class

**TEAE** treatment-emergent adverse event

triglycerides TG

WBC WHODrug do. **TSB** total serum bilirubin upper limit of normal white blood cell

World Health Organization Drug Dictionary

#### 1.0 **OBJECTIVES, ENDPOINTS AND ESTIMANDS**

#### 1.1 **Objectives**

#### 1.1.1 **Primary Objective**

- To evaluate the efficacy of TAK-625 in the primary cohort.
- To evaluate the safety of TAK-625 in subjects with PFIC.

#### Secondary Objective(s) 1.1.2

- To evaluate the efficacy of TAK-625 in subjects with PFIC.
- To evaluate the PK of TAK-625 in subjects with PFIC.

#### 1.1.3 Additional Objective(s)

applicable Terms of Use applicable terms of the applic To evaluate primary, secondary, and exploratory endpoints in the supplemental cohort

#### 1.2 **Endpoints**

#### 1.2.1 **Primary Endpoint(s)**

Change in the average morning ItchRO (Obs) severity score between baseline and average of Week 15 through Week 26.

#### 1.2.2 Secondary Endpoint(s)

#### 1.2.2.1 *Key Secondary Endpoints(s)*

- Change in the average morning ItchRO (Obs) frequency score between baseline and average of Week 15 through Week 26.
- Change in total sBA between baseline and Week 26

### 1.2.2.2 Secondary Endpoint(s)

- Proportion of subjects who experience an sBA control (defined as a reduction to <102 $\mu$ mol/L, or a reduction of >75%, or normalization) from baseline through Week 26.
- Change in the ItchRO (Obs) weekly average severity (based on daily maximum of morning and evening severity scores) between baseline and average of Week 15 through Week 26.



# 1.2.4 Safety Endpoints

• Incidence of AEs including SAEs, related to study drug, leading to study drug discontinuation, and AEs of clinical interest (AECIs).

AECIs include the following:

- LSV deficiency events.
- Liver parameter disruption.
- ns of Use Change from baseline in clinical laboratory values (hematology, chemistry, urinalysis, and others), physical examination findings (including body weight, height, and body mass index [BMI]), vital signs, and electrocardiogram (ECG) parameters

#### 1.2.5 **Other Endpoints**

#### 1.2.5.1 PK Endpoint

- Plasma levels of TAK-625 at predose and approximately 2.5 hours after the morning dose at Week 10.
- Plasma levels of TAK-625 at predose (optional) and approximately 30 minutes after morning dose at Week 14 (or any visit up to Week 26).

#### 1.3 Estimand(s)

Not Applicable.

#### 2.0 STUDY DESIGN

This is a phase 3, multicenter, open-label, uncontrolled study to evaluate the efficacy and safety of TAK-625 in the treatment of Japanese subjects with PFIC. Study Population:

The study population is defined as Japanese patients with PFIC who are 1 year of age or older". Subjects diagnosed with PFIC2 due to ABCB11 mutation that predicts residual BSEP function (nt-PFIC2) will be enrolled in the primary cohort. Subjects with other PFIC subtypes (eg, t-PFIC2, PFIC1/3/4 or other PFIC mutation variants) or postsurgical subjects (eg, internal or external biliary diversion surgery) will be enrolled in the supplemental cohort. (Subjects diagnosed with PFIC2 due to ABCB11 mutation that predicts complete absence of BSEP function [t-PFIC2] are excluded from the primary cohort and can be enrolled only in the supplemental cohort. PFIC subtypes should be determined by a genotyping [refer to Protocol Section 7.11).

Study Period (Screening, Treatment [Dose Escalation, Stable Dosing, and Follow-Up Dosing], and Safety Follow-Up Period):

This study consists of the screening period (up to 6 weeks prior to the study administration), 4-week dose escalation period (doses up to 600 µg/kg, BID, as tolerated), 44-week stable dosing period, and follow-up dosing period (until TAK-625 is approved or available in Japan commercially, or if the subject withdraws from the study, or if the investigator determines the subject's discontinuation, or if the sponsor stops the program or development in this indication).

### 1. Screening Period (up to 6 Weeks prior to the Study Administration):

In the screening period, for subjects who do not have documentation of mutation related with PFIC, a blood sample will be obtained for genotyping. Subjects diagnosed with PFIC2 (nt-PFIC2) will be enrolled in the primary cohort and those with other types of PFIC will be enrolled in the supplemental cohort. The electronic Diary (eDiary) for assessing pruritus with the Itch Reported Outcome (ItchRO) instrument will be dispensed and subjects and caregivers will undergo training during the screening visit.

### 2. Dose Escalation Period (4 weeks [up to 6 weeks]: Week 0 to 4 [6]):

In the dose escalation period, at the baseline visit (Week 0/Visit 2), subjects will be assessed to confirm continued study eligibility and undergo a physical examination including body weight, height, BMI, and vital signs, and have urine and blood samples taken for hematology, chemistry, fasting lipid panel, baseline levels of sBA and other cholestasis biochemical markers. Compliance with ItchRO will be assessed. Study drug will be supplied at each visit (Week 0/Visit 2, Week 2/Visit 3, and Week 4/Visit 4). The subject contacts (phone calls) will be conducted at Weeks 1 and 3. The dose is increased weekly, 150 µg/kg, 300 µg/kg, 450 µg/kg, and 600 µg/kg, BID.

Dose escalation should occur in the absence of major safety (eg, liver parameters and LSV deficiency) or tolerability concerns (eg, GI-related TEAEs) related or possibly related to study drug. Subjects with such safety concerns can be down-titrated to a lower, previously tolerated dose level for 1 week before continuing dose escalation. The minimum dose to continue in the study will be  $150 \, \mu \text{g/kg}$ , BID; subjects who cannot tolerate this dose will be discontinued from the study. The dose escalation period is allowed to be extended up to 6 weeks depending on the safety or tolerability concerns (refer to Protocol Section 8.1.3).

### 3. Stable Dosing Period (44 weeks: Week 5 to 48):

After the dose escalation period, each subject will continue dosing with study drug at the Week 4 or Week 6 dose level (the maximum tolerated dose [MTD] level) in the stable dosing period. Subjects will return to the study site at Weeks 6, 10, 14, 18, 22, 26, 28, 32, 36, 40, 44, and 48 and undergo physical examinations. Subject contacts (phone calls) will be conducted as appropriate throughout the stable dosing period. Subjects and caregivers will continue twice daily completion of their ItchRO throughout the period.

### 4. Follow-up Dosing Period (after Week 48):

Additionally, in the follow-up dosing period, each subject will continue dosing with study drug. The safety evaluation will be performed in all the subjects every 12 weeks from Week 48 visit until TAK-625 is approved or available in Japan commercially, or if the subject withdraws from the study, or if the investigator determines the subject's discontinuation, or if the sponsor stops the program or development in this indication. Bile acids and ItchRO will be measured to evaluate the long-term effectiveness of TAK-625. For subjects discontinuing early, safety follow-up will be conducted.

### 5. Safety Follow-up (after Final Visit/ET):

Subjects/caregivers will have a final safety follow-up subject contact (phone call) 7 days after the final study visit or ET visit (except for screen failure).

A schematic of the study design is included as Figure 2.a. A schedule of assessments is listed in Protocol Appendix A.

Figure 2.a **Schematic Study Design** 



ID=twice daily, SCR=screening, W=week, wks=weeks

#### 3.0 STATISTICAL HYPOTHESES AND DECISION RULES

Not Applicable.

### SAMPLE-SIZE DETERMINATION 4.0

PFIC is a rare disease. The targeted sample size of the primary cohort is approximately 3 subjects, and that of the supplemental cohort is approximately 6 subjects, based on enrollment feasibility of this population in Japan, rather than power calculation.

### ANALYSIS SETS

# All subjects who signed the informed consent form. All Subjects Who Signed the Informed Consent Form

#### 5.2 All Subjects Who Did Not Enter the Treatment Period

All subjects who did not enter the treatment period.

#### 5.3 Safety Analysis Set

All subjects who received at least one dose of study drug.

#### 5.4 **Intention-to-treat set (ITT)**

All subjects who received at least one dose of study drug.

#### 5.5 **Per-Protocol Analysis Set (PPS)**

ble Lekins of Use All ITT subjects who did not have any of the following major protocol deviations and whose primary endpoint was evaluable.

- Subjects who did not meet inclusion criteria #3, 4, 5, 6.
- Subjects who met exclusion criteria #1,2, 3, 4, 5, 6, 7, 9, 15, 16, 17, 19

#### STATISTICAL ANALYSIS 6.0

#### 6.1 **General Considerations**

The following definitions and calculation formulas will be used.

- Treatment-emergent adverse event (TEAE): An adverse event whose date of onset occurs on or after the start of study drug.
- Pretreatment event (PTE): Any untoward medical occurrence in a clinical investigation subject who has signed informed consent to participate in a study but prior to administration of study drug.
- Descriptive statistics for endpoints: Number of subjects, mean, standard deviation, standard error, maximum, minimum, and quartiles (Q1, median, and Q3).
- Duration of exposure to study drug (days): {Date of last dose of study drug date of first dose of study drug +1.
- Duration of study after baseline (days): {Date of last visit/contact date of first dose of study drug \ \P.
- Study drug compliance (%): Number of study drugs taken / (duration of exposure to study drug \*2) \* 100 (rounded to 1 decimal place).
- Dose Level (µg/kg): Strength of study drug taken (mg) / (last available body weight (kg) prior to or on the day of study drug taken) \* 1000.
  - Total Drug Exposure (μg/kg): Sum of {number of study drugs taken \* dose level received
- Average Daily Dose (µg/kg/day): Total Drug Exposure (µg/kg) / Duration of exposure to study drug (days).
- ItchRO (Obs/Pt) Daily Maximum of Morning and Evening Scores: Maximum of morning and evening severity scores for each day. The morning and evening severity scores CONFIDENTIAL

of the same day should be used for the calculation. Both the morning and evening ItchRO reports have a minimum score of 0 and a maximum score of 4, with 4 representing more severe (Item 1) itching.

- **Time to liver-associated events**: PEBD surgery, listing for liver transplantation, liver decompensation [hepatic encephalopathy, variceal bleeding, ascites, and spontaneous bacterial peritonitis] events, hepatocellular carcinoma (HCC), death, and other.
- Estimated Total Lipids (mg/dL): Cholesterol (mg/dL) + Triglycerides (mg/dL)
- Ratio of Alpha-tocopherol to Estimated Total Lipids (mg/g): 1000 \* Alpha-tocopherol (mg/dL) / Estimated Total Lipids (mg/dL). For Alpha-tocopherol concentrations reported as below the minimum quantitation limit, half of the minimum quantitation limit is used in the calculation.
- Corrected Sodium (mEq/L): sodium (mEq/L) + (0.002 \* Triglycerides (mg/dL)).
- FIB-4: (Age (years) \* AST (U/L)) / (platelet count (10^9/L) \* sqrt(ALT(U/L)))
  - Age (years) is years at sample collection visit.
- APRI:  $100 * (AST (U/L) / AST ULN(U/L)) / (platelet count (10^9/L))$ 
  - > ULN is upper limit normal
- **Significant Protocol Deviation**: Deviation defined in the PDMP as "Important PD" whose Severity Classifications is "major" or "critical".
- Time since original diagnosis of PFIC (months): (date of first dose date of original diagnosis of PFIC + 1) / 30.4375.

When reporting derived values or parameters, following presenting rules will be applied.

- For sBA, ItchRO: For rules on rounding and decimal presentation of these statistics, along with the rules for presenting certain derived values see below.
  - For measures of median and mean, use 3 decimal places.
  - For measures of standard deviation, standard error of the mean and CI, use 4 decimal places.
  - For measures of minimum and maximum values as well as observed value (for Listing), use 2 decimal places.
  - >=5 is rounded up away from zero, whereas <5 is rounded down toward zero, to account for rounding of negative numbers.
  - For p-values use 3 decimal places.
  - Presentation of p-values display p-values that would round to 0.000 as <0.001.
- Other than sBA, and ItchRO: For rules on rounding and decimal presentation of these statistics, along with the rules for presenting certain derived values see below.

- For measures of median and mean, use 1 decimal place beyond those used for the measurement.
- For measures of standard deviation, standard error of the mean and CI, use 2 decimal places beyond those used for the measurement.
- For measures of minimum and maximum values, use the same number of decimal places as those used for the measurement.
- >=5 is rounded up away from zero, whereas <5 is rounded down toward zero, to account for rounding of negative numbers.
- For p-values use 3 decimal places.
- > Presentation of p-values display p-values that would round to 0.000 as <0.001.
- > BMI should be rounded to 1 decimal place for reporting.
- ➤ Derived questionnaire scores, and other similar efficacy parameters recorded as integers, should be rounded to 1 decimal place for reporting.
- Averaged lab results (e.g. Diastolic/Systolic Blood Pressure and Pulse [when taken in triplicate]) should be rounded to 1 decimal place for reporting.

### 6.2 Analysis Approach

### **6.2.1** Analysis Cohort

Analyses described in section  $6.3 \sim 6.8$  will be performed for primary cohort.

### 6.2.2 Analysis Approach for Continuous Efficacy Endpoints

For efficacy endpoints, all continuous endpoints in this trial will use the analysis method below unless stated otherwise in the section specific to an endpoint.

 Descriptive statistics and two-sided 95% confidence interval of mean will be provided for observed values (baseline and post-baseline visits) and changes from baseline (each postbaseline visit - baseline). For endpoint with multiple visits, these will be provided by visit.

### 6.2.3 Analysis Approach for Binary Efficacy Endpoints

For efficacy endpoints, all binary endpoints in this trial will use the analysis method below unless stated otherwise in the section specific to an endpoint.

Frequency distribution will be provided by visit, with proportion and the two-sided 95% confidence interval. For endpoint with multiple visits, these will be provided by visit.

### 6.2.4 Analysis Approach for Time-to-Event Efficacy Endpoints

For efficacy endpoints, all time-to-event endpoints in this study will use the analysis method below unless stated otherwise in the section specific to an endpoint.

The event-free survival rate and the two-sided 95% confidence intervals will be provided using the Kaplan-Meier method. The event-free survival rate will also be plotted. Time to event will be defined as the date of first dose of study drug to the event which comes fastest. For subjects without an event, time to event will be defined as the date of first dose of Lekk study drug to the censoring date, which is the date of the last study visit/contact.

#### 6.3 **Disposition of Subjects**

#### 6.3.1 **Study Information**

All Subjects Who Signed the Informed Consent Form

Date First Subject Signed Informed Consent F

Date of Last Subject Analysis Set:

Analysis Endpoint(s):

MedDRA Dictionary Version

WHO Drug Dictionary Version

SAS Version Used for Creating the Datasets

(1) Study Information Analytical Method(s):

Study information shown in the analysis endpoints section will be

provided.

6.3.2 **Disposition of Subjects** 

Analysis Set:

Study Drug Completion Analysis Endpoint(s): [Completed Study Drug, Prematurely

> Status Discontinued Study Drug

Reason for Discontinuation [AE, Protocol Deviation, Lost to

of Study Drug Follow-up, Withdrawal by Subject, Study Terminated by Sponsor,

Pregnancy, Lack of Efficacy, Other]

Completion Status of All [Completed Study, Prematurely

Planned Study Visits Discontinued Study]

Reason for Discontinuation [AE, Protocol Deviation, Lost to Follow-up, Withdrawal by Subject, of Study

Study Terminated by Sponsor, Pregnancy, Lack of Efficacy, Other]

Property of Lakega: For no, (1) Disposition of Subjects

Frequency distributions will be provided. When calculating

percentages for the reasons for discontinuation, the total number of

subjects who prematurely discontinued will be used as the denominator.

#### 6.3.3 **Protocol Deviations and Analysis Sets**

#### 6.3.3.1 Significant Protocol Deviations

Analysis Set: ITT

Significant Protocol Deviation [Informed Consent and Process, Analysis Endpoint(s):

> Inclusion Criteria, Exclusion Criteria, Concomitant Medication, Laboratory Assessment, Study Procedures (not safety and efficacy related), Safety, Visit Schedule, IP conditions, IP preparation, IP administration, Subject IP Compliance, Efficacy,

Subject Discontinuation,

Administrative, Patient Reported Outcomes, PK/PD, Other Criteria]

Analytical Method(s): (1) Protocol Deviations

> Frequency distribution will be provided for each deviation category. A subject who has several deviations will be counted once in each appropriate category. A subject who has several deviations that can be

classified into the same category will be counted only once.

6.3.3.2 Analysis Sets

Analysis Endpoint(s). Property of Takeda.

Handling of Subjects [Categories are based on the definitions in

Section 5.0]

**Analysis Sets** 

ITT [Included]

**PPS** [Included]

Safety Analysis Set [Included]

Analytical Method(s): (1) Subjects Excluded from Analysis Sets

(2) Analysis Sets

Frequency distributions will be provided. For (1), a subject who has several reasons for exclusion will be counted once in each appropriate

CONFIDENTIAL

Who Leiths of Use category. A subject who has several reasons for exclusion that can be classified into the same category will be counted only once.

#### 6.4 **Concomitant Medications**

Analysis Set: ITT

Analysis Endpoint(s): **Concomitant Medications** 

(1) Concomitant Medications That Started Prior to and Were Ongoing Analytical Method(s):

at Baseline as well as Those That Started After Baseline by Anatomical Therapeutic Chemical Level 2 and Preferred

Medication Name

Frequency distributions will be provided. WHO Drug dictionary will be used for coding. Summaries will be provided using anatomical therapeutic chemical level 2 and preferred medication names and sorted in decreasing frequency based on the number of reports. A subject who has been administered several medications with the same preferred medication names will be counted only once for that preferred medication names. For anatomical therapeutic chemical anner.

Anner.

Anner. level 2, same manners in counting frequency.

### **6.5** Extent of Exposure and Compliance

Analysis Set: ITT

Analysis Endpoint(s): Duration of Exposure to  $[0 \le - \le 28, 29 \le - \le Max]$ 

Study Drug (days)

Study Drug Compliance (%) [Min<= - < 80, 80 <= - <= 100, 100< -

 $\leq=Max$ 

Total Drug Exposure (µg/kg)

Average Daily Dose

(µg/kg/day)

Analytical Method(s): (1) Study Drug Exposure, Compliance, Total Drug Exposure and

Average Daily Dose

Frequency distributions for categorical endpoints and descriptive

statistics for continuous endpoints will be provided.

### 6.6 Efficacy Analysis







#### 6.7 **Safety Analysis**

#### 6.7.1 **Adverse Events**

6.7.1.1 Overview of Treatment-Emergent Adverse Events

Analysis Set: Safety Analysis Set

Analysis Endpoint(s): TEAE

[Related, Not Related] Categories: Relationship to Study Drug

> [Mild, Moderate, Severe] Intensity

The following summaries will be provided. Analytical Method(s):

(1) Overview of Treatment-Emergent Adverse Events

- 1) All Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
- 2) Relationship of Treatment-Emergent Adverse Events to study drug (number of events, number and percentage of subjects)
- 3) Intensity of Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
- 4) Treatment Emergent Adverse Events leading to study drug discontinuation (number of events, number and percentage of subjects)
- 5) Serious Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
- Relationship of serious Treatment-Emergent Adverse Events to study drug (number of events, number and percentage of subjects)
- 7) Serious Treatment-Emergent Adverse Events leading to study drug discontinuation (number of events, number and percentage of subjects)
- Property of Takeda. For non-8) Treatment-Emergent Adverse Events resulting in death (number of events, number and percentage of subjects)

TEAEs will be counted according to the rules below.

### Number of subjects

- Summaries for 2) and 6) A subject with occurrences of TEAE in both categories (i.e., Related and Not Related) will be counted once in the Related category.
- Summary for 3) A subject with multiple occurrences of TEAE will be counted once for the TEAE with the maximum intensity,
- Summaries other than 2), 3), and 6) A subject with multiple occurrences of TEAE will be counted only once.

### Number of events

For each summary, the total number of events will be calculated.

### 6.7.1.2 Displays of Treatment-Emergent Adverse events

Safety Analysis Set Analysis Set:

**TEAE** Analysis Endpoint(s):

Categories: Intensity [Mild, Moderate, Severe]

> Time of Onset (day) [1-28, 29-197, 198-336, 337-

> > Max

Analytical Method(s): The following summaries will be provided using frequency Property of Takeda. For not distribution.

TEAEs will be coded using the MedDRA and will be summarized using SOC and PT.

SOC will be sorted alphabetically and PT will be sorted in decreasing frequency for tables provided by SOC and PT. SOC and PT will be sorted in decreasing frequency for tables provided by System Organ Class only or PT only.

- (1) Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (2) Treatment-Emergent Adverse Events by System Organ Class
- (3) Treatment-Emergent Adverse Events by Preferred Term
- (4) Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term

- (6) Intensity of Drug-Related Treatment-Emergent Adverse Events by System Organ Class, and Preferred Term

  (7) Treatment-Emergent Adverse Events Leading to Study B Discontinuation by System
- (8) Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (9) Treatment-Emergent Adverse Events by System Organ Class and Preferred Term Over Time
- Treatment-Emergent Adverse Events of Clinical Interest by (10)System Organ Class and Preferred Term
- Drug-Related Treatment-Emergent Adverse Events of Clinical Interest by System Organ Class and Preferred Term

The frequency distribution will be provided according to the rules below.

### Number of subjects

- Summary tables other than (5), (6) and (9) A subject with multiple occurrences of TEAE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of TEAE within a PT will be counted only once in that PT. Percentages will be based on the number of subjects in the safety analysis set.
- Summary tables for (5) and (6) A subject with multiple occurrences of TEAE within a SOC or a PT will be counted only once for the TEAE with the maximum intensity. Percentages will be based on the number of subjects in the safety analysis set.
- Property of Takeda. For none Summary table for (9) A subject with a TEAE that occurs in more than one interval is counted in all the intervals that the TEAE occurs. For each time interval, a subject with multiple occurrences of TEAE within a SOC or a PT will be counted only once in that SOC or PT. When calculating percentages for each time interval, the number of subjects at risk (i.e., subjects who either have an exposure or have an occurrence of TEAE, during or after the corresponding time interval) will be used as the denominator. The number of

cable Terms of Use subjects whose onset of any one of the TEAEs is within the time interval will be used as the numerator.

#### 6.7.2 **Clinical Laboratory Evaluations**

6.7.2.1 Laboratory Tests other than Urinalysis

Analysis Set: Safety Analysis Set Analysis Endpoint(s): See Section 9.3.6.

Using the visits (Baseline to post Baseline visits) of the visit window Visit:

defined in Section 9.2.2.

For each endpoint, summaries (1) to (3) will be provided. Analytical Method(s):

(1) Summary of Laboratory Test Results and Change from Baseline

by Visit

Descriptive statistics for observed values and changes from baseline (each post-baseline visit - Baseline) will be provided for

each visit.

(2) Case Plots

Plots over time for each subject will be presented.

(3) Summary of Shifts of Laboratory Test Results Shift tables showing the number of subjects in each category at

baseline and each post-baseline visit will be provided.

For each laboratory test, the laboratory values will be classified as "Low", "Normal" or "High" relative to the normal reference range provided by the central laboratory. The shift tables will be based

on these classifications.

### Urinalysis 6.7.2.2

Analysis Set: Safety Analysis Set

Analysis Endpoint(s): See Section 9.3.6.

Analytical Method(s): Using the visits (Baseline to post Baseline visits) of the visit window

defined in Section 9.2.2.

For pH and specific gravity, summaries (1), (2) and (4) will be

provided.

For each endpoint other than pH and specific gravity, summaries (3)

and (4) will be provided.

(1) Summary of Urine Laboratory Test Results and Change from Baseline by Visit

### CONFIDENTIAL

Descriptive statistics for observed values and changes from baseline (each post-baseline visit - Baseline) will be provided for each visit.

(2) Case Plots Plots over time for each subject will be presented.

- (3) Number of Subjects in Categories of Urine Laboratory Test Results Shift tables showing the number of subjects in each category at baseline and each post-baseline visit will be provided.
- (4) Summary of Shifts of Urine Laboratory Test Results Shift tables showing the number of subjects in each category at baseline and each post-baseline visit will be provided. For each urine laboratory test, the laboratory values will be classified as "Low", "Normal" or "High" relative to the normal reference range provided by the central laboratory. The shift tables will be based on these classifications.

#### 6.7.3 Vital Signs, Weight and Height

Safety Analysis Set Analysis Set:

Systolic Blood Pressure Analysis Endpoint(s): Diastolic Blood Pressure

> Heart Rate **Body Temperature**

Weight Height

Respiration Rate

Using the visits (Baseline to post Baseline visits) of the visit window Visit:

defined in Section 9.2.2.

Analytical Method(s): For each endpoint, summaries (1) and (2) will be provided. Property of Lakeda.

(1) Summary of Vital Signs, Weight and Height, and Change from Baseline by Visit Descriptive statistics for observed values and changes from baseline (each post-baseline visit - Baseline) will be provided for each visit.

(2) Case Plots

Plots over time for each subject will be presented.

#### 6.7.4 **ECGs**

Safety Analysis Set Analysis Set:

Analysis Endpoint(s): Heart Rate

> RR Interval PR Interval **QRS** Interval QT Interval QTcF Interval

[Within Normal Limits, Abnormal but not Interpretation

Clinically Significant, Abnormal and

Clinically Significant]

Using the visits (Baseline to post Baseline visits) of the visit window Visit:

defined in Section 9.2.2.

For each endpoint other than 12-lead ECG interpretations, summaries Analytical Method(s):

(1) and (2) will be provided.

For ECG interpretation, summary (3) will be provided.

(1) Summary of EGG Parameters and Change from Baseline by Visit Descriptive statistics for observed values and changes from baseline (each post-baseline visit - Baseline) will be provided for each visit.

(2) Case Plots

Plots over time for each subject will be presented.

(3) Summary of Shift of ECG Interpretation Shift table showing the number of haseling. Shift table showing the number of subjects in each category at baseline and each post-baseline visit will be provided.

### Displays of Treatment-Emergent Adverse Events (Japanese) 6.7.5

Analysis Set: Safety Analysis Set

Analytical Method(s): **TEAE** 

TEAEs will be summarized in the same way as in Section 6.7.1.2. All

summaries will be presented in Japanese.

### 6.8 Pharmacokinetic, Pharmacodynamic, and Biomarker Analyses

### 6.8.1 Pharmacokinetic Analysis

Not applicable.

### 6.9 Other Analyses

### 6.9.1 Analyses for Overall Supplemental Cohort

Cohort: Overall Supplemental Cohort

Analytical Method(s): The same analyses in section  $6.3 \sim 6.8$  will be performed for overall

supplemental cohort.

### 6.9.2 Analyses for All Cohorts Combined

Cohort: All Cohorts Combined

Analytical Method(s): The same analyses in section 6.3 > 6.8 will be performed for all

cohorts combined.

### 7.0 REFERENCES

[1] World Health Organization (WHO) growth charts "A SAS Program for the WHO Growth Charts (ages 0 to < 2 years)" https://www.cdc.gov/nccdphp/dnpao/growthcharts/resources/sas-who.htm

[2] Centers for Disease Control (CDC) growth charts "A SAS Program for the 2000 CDC Growth Charts (ages 0 to < 20 years)" https://www.cdc.gov/nccdphp/dnpao/growthcharts/resources/sas.htm

### 8.0 CHANGES TO PROTOCOL PLANNED ANALYSES

There was no change to the protocol planned analyses.

### 9.0 APPENDIX

### 9.1 Changes From the Previous Version of the SAP

Not applicable.

### **9.2** Data Handling Conventions

### 9.2.1 Definition of Study Days

The following definitions and calculation formulas will be used.

• Study Day: The day before the first dose of the study drug will be defined as Study Day -1 and the day of the first dose will be defined as Study Day 1. If the date of the observation is

### CONFIDENTIAL

on the same date or after the day of the first dose, Study Day will be calculated relative to Study Day 1. Otherwise, Study Day will be calculated relative to Study Day -1.

 Follow-up Day: The day after the last dose of the study drug will be defined as Follow-up Day 1.

### 9.2.2 Definition of Study Visit Windows

When calculating Study Day relative to a reference date (i.e., date of first dose of study drug [Day 1]), if the date of the observation is on the same date or after the reference date, it will be calculated as: date of observation - reference date + 1; otherwise, it will be calculated as: date of observation - reference date. Hence, reference day is always Day 1 and there is no Day 0.

When calculating Follow-up Day relative to a reference date (i.e., date of last dose of study drug [Follow-up Day 0]), it will be calculated as: date of observation - reference date. Hence, reference day is always Follow-up Day 0.

All evaluable data (i.e., non-missing data) will be handled according to the following rules.

### 9.2.2.1 Endpoints other than ItchRO Scores and PK Samples

For each visit, observation obtained in the corresponding time interval will be used. If more than one observation lies within the same visit window, the observation with the closest Study Day to the scheduled Study Day will be used. If there are two observations equidistant to the scheduled Study Day, the later observation will be used. For laboratory test data, if there are two observations of both central laboratory sample and local sample on the same date, central laboratory sample data will be used. Values less than or equal to the lower limit of quantification will be treated as one-half of the lower limit value when calculating the descriptive statistics. Values greater than or equal to the upper limit of quantification will be treated as the upper limit value when calculating the descriptive statistics.

Table 9.1 Visit Window of sBA, sBA subspecies, C4, Serum Storage Sample

| Visit O | Scheduled Study Day<br>(days) | Time Interval (days) | |
|---|---|---|---|
| V 1511 | | Study Day | Follow-up Day |
| Baseline (Week 0) | Study Day: 1 | -42 - 1 | |
| Week 2 | Study Day: 15 | 2 - 29 | < 15 |
| Week 6 | Study Day: 43 | 30 - 57 | < 15 |
| Week 10 | Study Day: 71 | 58 - 85 | < 15 |
| Week 14 | Study Day: 99 | 86 - 113 | < 15 |
| Week 18 | Study Day: 127 | 114 - 141 | < 15 |

Table 9.1 Visit Window of sBA, sBA subspecies, C4, Serum Storage Sample

| Visit | Scheduled Study Day | Time Interval (days) | |
|---|---|---|---|
| VISIT | (days) | Study Day | Follow-up Dax |
| Week 22 | Study Day: 155 | 142 - 169 | < 15 |
| Week 26 | Study Day: 183 | 170 - 190 | 15 |
| Week 28 | Study Day: 197 | 191 - 211 | (15 × 15 |
| Week 32 | Study Day: 225 | 212 - 239 | < 15 |
| Week 36 | Study Day: 253 | 240 - 267 | < 15 |
| Week 40 | Study Day: 281 | 268 - 295 | < 15 |
| Week 44 | Study Day: 309 | 296 - 323 | < 15 |
| Week 48 | Study Day: 337 | 324 - 379 | < 15 |
| Week (48 + 12 * n) (n=1, 2, | 337 + 12 | (337 + 12 * 7 * | < 15 |
| ) | Study Day: $7 * (n)$ | (n) - 41) - (337 + | |
| | S | 12 * 7 * (n) + 42) | |

Table 9.2 Visit Window of Vital Signs, Weight and Height, for pruritus

Time Interval (days) Scheduled Study Day Visit (days) Study Day Follow-up Day Study Day: 1 Baseline (Week 0) -42 - 1 Study Day: 15 < 15 Week 2 2 - 22 Week 4 Study Day: 29 < 15 23 - 36Study Day: 43 Week 6 < 15 37 - 57 Study Day: 71 Week 10 < 15 58 - 85 Study Day: 99 Week 14 < 15 86 - 113 Study Day: 127 Week 18 < 15 114 - 141 Study Day: 155 Week 22 < 15 142 - 169

Table 9.2 Visit Window of Vital Signs, Weight and Height, for pruritus

| Visit | Scheduled Study Day | Time Interval (days) | |
|---|---|---|---|
| VISIT | (days) | Study Day | Follow-up Day |
| Week 26 | Study Day: 183 | 170 - 190 | <45 |
| Week 28 | Study Day: 197 | 191 - 211 | < 15 |
| Week 32 | Study Day: 225 | 212 - 239 | < 15 |
| Week 36 | Study Day: 253 | 240 - 26 | < 15 |
| Week 40 | Study Day: 281 | 268 - 295 | < 15 |
| Week 44 | Study Day: 309 | 296 - 323 | < 15 |
| Week 48 | Study Day: 337 | 324 - 379 | < 15 |
| Week (48 + 12 * n) (n=1, 2, | 337 + 12 | (337 + 12 * 7 * | < 15 |
| ) | Study Day: *7* (n) | (n) - 41) - (337 + | |
| | e e | 12 * 7 * (n) + 42) | |

Table 9.3 Urinalysis, Cholestasis Biomarkers (FGF19, Autotaxin)

| Visit | Scheduled Study Day | Time Interval (days) | |
|---|---|---|---|
| VISIT | (days) | Study Day | Follow-up Day |
| Baseline (Week 0) | Study Day: 1 | -42 - 1 | |
| Week 6 | Study Day: 43 | 2 - 57 | < 15 |
| Week 10 | Study Day: 71 | 58 - 99 | < 15 |
| Week 18 | Study Day: 127 | 100 - 155 | < 15 |
| Week 26 | Study Day: 183 | 156 – 197 | < 15 |
| Week 32 | Study Day: 225 | 198 - 253 | < 15 |
| Week 40 | Study Day: 281 | 254 - 309 | < 15 |
| Week 48 | Study Day: 337 | 310 - 379 | < 15 |

Urinalysis, Cholestasis Biomarkers (FGF19, Autotaxin) Table 9.3

| Visit | Scheduled Study Day | Time Interval (days) | |
|---|---|---|---|
| VISIT | (days) | Study Day | Follow-up Dax |
| Week (48 + 12 * n) (n=1, 2, | 337 + 12 | (337 + 12 * 7 * | < 15 |
| ) | Study Day: ${337 + 12 \atop *7*(n)}$ | (n) - 41) - (337 + | 2/0 |
| | , , | 12 * 7 * (n) + 42) | .: 00. |

Table 9.4 Lipid Panel, Lipid Soluble Vitamins

| | | 12 * 7 * (n) + 42) | |
|---|---|---|---|
| Table 9.4 Lipid Panel, L | ipid Soluble Vitamins | No of | ppli |
| Visit | Scheduled Study Day | Time Inter | val (days) |
| VISIt | (days) | Study Day | Follow-up Day |
| Baseline (Week 0) | Study Day: 1 | -42 – 1 | |
| Week 6 | Study Day: 43 | 2 – 57 | < 15 |
| Week 10 | Study Day: 71 | 58 – 85 | < 15 |
| Week 14 | Study Day: 99 | 86 – 113 | < 15 |
| Week 18 | Study Day: 127 | 114 – 141 | < 15 |
| Week 22 | Study Day: 155 | 142 – 169 | < 15 |
| Week 26 | Study Day: 183 | 170 – 197 | < 15 |
| Week 32 | Study Day: 225 | 198 - 253 | < 15 |
| Week 40 | Study Day: 281 | 254 - 309 | < 15 |
| Week 48 | Study Day: 337 | 310 - 379 | < 15 |
| Week (48 + 12 * n) (n=1, 2, | Star In Day 337 + 12 | (337 + 12 * 7 * | < 15 |
| Week (48 + 42 * n) (n=1, 2,) | Study Day: ${}^{337+12}_{*7*(n)}$ | (n) - 41) - (337 + | |
| C 1.0 | | 12 * 7 * (n) + 42) | |

Table 9.5 CBC, Coagulation, Chemistry Panel

| Visit | Scheduled Study Day | Time Interval (days) | |
|---|---|---|---|
| VISIt | (days) | Study Day | Follow-up Day |
| Baseline (Week 0) | Study Day: 1 | -42 - 1 | 101 |
| Week 2 | Study Day: 15 | 2 - 29 | 15 |
| Week 6 | Study Day: 43 | 30 - 57 | (15 × 15 |
| Week 10 | Study Day: 71 | 58 - 85 | < 15 |
| Week 14 | Study Day: 99 | 86 - H3 | < 15 |
| Week 18 | Study Day: 127 | 144 - 141 | < 15 |
| Week 22 | Study Day: 155 | 142 - 169 | < 15 |
| Week 26 | Study Day: 183 | 170 - 197 | < 15 |
| Week 32 | Study Day: 225 | 198 - 253 | < 15 |
| Week 40 | Study Day: 281 | 254 - 309 | < 15 |
| Week 48 | Study Day: 337 | 310 - 379 | < 15 |
| Week (48 + 12 * n) (n=1, 2, | 337 + 12 | (337 + 12 * 7 * | < 15 |
| ) | Study Day: *7 * (n) | (n) - 41) - (337 + | |
| | | 12 * 7 * (n) + 42) | |

Table 9.6 Visit Window of ECGs, AFP

| Visit | Scheduled Study Day<br>(days) | Time Interval (days) | |
|---|---|---|---|
| Visit | | Study Day | Follow-up Day |
| Baseline (Week 0) | Study Day: 1 | -42 - 1 | |
| Week 10 | Study Day: 71 | 2 - 127 | < 15 |
| Week 26 | Study Day: 183 | 128 - 197 | < 15 |
| Week 48 | Study Day: 337 | 198 - 379 | < 15 |

Table 9.6 Visit Window of ECGs, AFP

| Visit | Scheduled Study Day | Time Interval (days) | |
|---|---|---|---|
| V 151t | (days) | Study Day | Follow-up Dax |
| Week (48 + 12 * n) (n=1, 2, | 337 + 12 | (337 + 12 * 7 * | < 15 |
| ) | Study Day: ${337 + 12 \atop *7 * (n)}$ | (n) - 41) - (337 + | 2/0 |
| | , , | 12 * 7 * (n) + 42) | 03. |



Average ItchRO Scores

For each visit other than Week 6, average ItchRO score is defined as the average of the scores (morning, evening, or daily maximum of morning and evening) over the visit consisting of the 28 days on or before the scheduled Study Day (i.e., the sum of the score) of non-missing scores). The answer "I don't know"

For Week 6 average ItchRO score is defined as the average of the score (morning, evening, or daily maximum of morning and evening) over the visit consisting of the score of non-missing scores).

For Week 6, average ItchRO score is defined as the average of the scores (morning, evening, or daily maximum of morning and evening) over the visit consisting of the 41 days on or before the scheduled Study Day (i.e., the sum of the scores divided by the number of non-missing scores). The answer "I don't know" will be treated as missing.

In the event that a subject/caregiver failed to complete the morning/evening report, the morning/evening score for that day will be treated as missing data. If 25% or more ItchRO scores A sich Rerage Ity and and see only and are reage Ity and are represented the commercial use only and are represented to the reage Ity and are represented to the reage Ity and are represented to the reage Ity and are reage Ity an for the post-baseline visit are missing, the average ItchRO score at that visit will be treated as missing. The restriction is not set for baseline average ItchRO scores.
Table 9.8 Visit Window of Average ItchRO Score

| Visit | Scheduled Study Day | Time Inter | val (days) |
|---|---|---|---|
| V 151t | (days) | Study Day | Follow-up Day |
| Baseline (Week 0) | Study Day: -1 | -281 | 10 |
| Week 6 | Study Day: 42 | 2 - 42 | S 15 |
| Week 10 | Study Day: 70 | 43 - 70 | < 15 |
| Week 14 | Study Day: 98 | 71 - 98 | < 15 |
| Week 18 | Study Day: 126 | 99 - 126 | < 15 |
| Week 22 | Study Day: 154 | 127 - 154 | < 15 |
| Week 26 | Study Day: 182 | 155 - 182 | < 15 |
| Week 28 | Study Day: 197 | 170 - 197 | < 15 |
| Week 32 | Study Day: 225 | 198 - 225 | < 15 |
| Week 36 | Study Day: 253 | 226 - 253 | < 15 |
| Week 40 | Study Day: 281 | 254 - 281 | < 15 |
| Week 44 | Study Day: 309 | 282 - 309 | < 15 |
| Week 48 | Study Day: 337 | 310 - 337 | < 15 |
| Week (48 + 12 * n) (n=1,2, | St. 1 D 337 + 12 | (337 + 12 * 7 * | < 15 |
| ) ,011 | Study Day: * 7 * (n) | (n) - 27) - (337 + | |
| | | 12 * 7 * (n) | |

# 9.2.3 Partial Date Conventions

For Medication History and Concomitant Medication, if their stop date is partially/completely missing, following handling rules will be applied.

```
if (CMCAT="MEDICATION HISTORY") then "(1) Medical History "; else if (CMENRTPT="ONGOING") then "(3) Concomitant Medication"; else if
```

( . < medication end year < TAK-625 start year) or ( medication end year = TAK-625 start year and

CONFIDENTIAL

```
. < medication end month < TAK-625 start month) or

( medication end year = TAK-625 start year and medication end month = TAK-625 start month and . < medication end date < TAK-625 start date ) then "(2) Concomitant Medication"; else "(3) Concomitant Medication";
```

# 9.3 Derivation of Endpoints

# 9.3.1 Primary Efficacy Endpoints

Both the morning and evening ItchRO reports have a minimum score of 0 and a maximum score of 4, with 4 representing more severe (Item 1) itching. The derivation method for the primary efficacy endpoint will be described below.

After the derivation described in section 9.2.2.3, each subject will have a baseline (Week 0) average morning ItchRO (Obs) severity score, and have post-baseline average morning ItchRO (Obs) severity scores at Weeks 18, Week 22, and Week 26. For each subject, change in the average morning ItchRO (Obs) severity score between baseline and post-baseline visit can be calculated at Weeks 18, Week 22, and Week 26. Hence, the primary efficacy endpoint for each subject can be calculated as an average of the changes in the average morning ItchRO (Obs) severity score from Week 15 through Week 26 (i.e., the sum of the average morning ItchRO (Obs) severity scores divided by the number of non-missing morning severity scores).

# 9.3.2 Average ItchRO Scores

For ItchRO scores, both the morning and evening ItchRO reports have a minimum score of 0 and a maximum score of 4, with 4 representing more severe (Item 1) or more frequent (Item 3) itching. After the derivation described in section 9.2.2.3, the following endpoints will be derived the same procedures as section 9.3.1.



• Change in the average evening ItchRO (Obs/Pt) severity score between baseline and average of Week 15 through Week 26.

- Change in the average ItchRO (Obs/Pt) severity and frequency (based on daily maximum of morning and evening severity scores) between baseline and average of Week 15 through Week 26.
- Change in the average morning ItchRO (Obs/Pt) frequency score between baseline and average of Week 15 through Week 26.
- Change in the average evening ItchRO (Obs/Pt) frequency score between baseline and average of Week 15 through Week 26.

# 9.3.3 Responder Endpoints

• Subjects who experience an sBA control: subjects with a reduction to  $<102 \mu Mol/L$ , or a reduction of >75%, or normalization) from baseline through Week 26





# **9.3.5 Z-scores**

Z-scores of weight, height and BMI are based on a subject's gender and age at each scheduled visit. For subjects less than 24 months of age, the World Health Organization (WHO) growth charts are recommended by the Centers for Disease Control (CDC) and will be used to derive z-scores. For subjects at least 24 months of age, the CDC growth charts will be used to derive z-scores.

Age at which height and weight were measured should be used for calculating z-scores, not using age at baseline.

# 9.3.6 Lists of Laboratory Tests

| | | •,0 | |
|---|---|---|---|
| Hematology (CBC with | <b>Chemistry</b> | Lipid Panel | <u>Urinalysis</u> |
| <u>Differential</u> ) | Albumin | Total cholesterol | pH |
| Hematocrit | ALP | LDL-C (direct) | Specific gravity |
| Hemoglobin | Amylase | HDL-C | Protein |
| MCV, MCH, MCHC | ALT (SGPT) | TG | Glucose |
| Red blood cells | AST (SGOT) | ), | Ketones |
| Platelets | Bicarbonate | <b>Cholestasis Biomarkers</b> | Bilirubin |
| White blood cells | Bilirubin, direct | sBA (LC-MS) | Occult blood and cells |
| WBC Differential (% and | (conjugated) | sBA subspecies | Nitrite |
| absolute) | TSB | 7alpha-hydroxy-4- | Urobilinogen |
| Neutrophils | BUN | cholesten-3-one (C4) | Leukocyte esterase |
| Eosinophils | Calcium | FGF-19 | Microscopic examination |
| Basophils | Chloride | Autotaxin | Oxalate |
| Lymphocytes | Creatinine | | Urinary creatinine |
| Monocytes | GGT | Lipid Soluble | J |
| ₹0. | Glucose | <u>Vitamins</u> | Marker of HCC |
| <b>Coagulation</b> | Lipase | 25-hydroxy vitamin D | AFP* |
| aPTT (sec) | Phosphate | Retinol | |
| INR | Potassium | RBP | |
| PT (sec) | Sodium | Alpha-tocopherol | |
| 0, | Corrected Sodium | Estimated Total Lipids | |
| | Total protein | Ratio of Alpha-tocopherol | |
| | Total sBA (enzymatic assay) | to Estimated Total Lipids | |
| | Uric Acid | | |
| | Measured serum<br>Osmolality | | |

# Property of Takeda: For non commercial use only and subject to the applicable Terms of tuse

Properly of Takeda: For non-commercial use only and subject to the applicable Terms



# STATISTICAL ANALYSIS PLAN for Week 26

Study Number: TAK-625-3002

applicable Terms of Use A J-3002

Attack the Effica

Assive Familial Intra

Phase: 3

Version: 2.0

Date: 10-Nov-2023

ased on:

Protocol Version: Amendment 2

Protocol Date: 08-Dec-2022 Study Title: An Open-Label, Phase 3 Study to Evaluate the Efficacy and Safety of TAK-625 in the Treatment of Subjects with Progressive Familial Intrahepatic Cholestasis

Jn:
Arotocol Version: Amendma
Protocol Date: 08-Dec-2022

| | Approval Date | Primary Rationale for Revision |
|---|---|---|
| 1.0 | 01-Jul-2022 | Primary Rationale for Revision Not Applicable |
| 2.0 | | See Section 9.1 |
| | | Not Applicable See Section 9.1 Primary Rationale for Revision Not Applicable See Section 9.1 Applicable Terror Te |
| | | Niectxo |
| | | Mandsv |
| | | ial use of |
| | contine | |
| <b>.</b> | ornon | |
| Lego. | | |
| 10 | | |
| of San | | |

# TABLE OF CONTENTS

| 1.0 | OBJEC | CTIVES, ENDPOINTS AND ESTIMANDS | 9 |
|---|---|---|---|
| 1. | 1 Ob | jectives | |
| | 1.1.1 | Primary Objective | 9 |
| | 1.1.2 | Secondary Objective(s) | <b>.(.)</b> 9 |
| | 1.1.3 | Additional Objective(s) | 9 |
| 1.2 | 2 End | dpoints | 9 |
| | 1.2.1 | Additional Objective(s) dpoints Primary Endpoint(s) Secondary Endpoint(s) .2.1 Key Secondary Endpoints(s) | 9 |
| | 1.2.2 | Secondary Endpoint(s) | 9 |
| | 1.2 | .2.1 Key Secondary Endpoints(s) | 9 |
| | 1.2 | .2.2 Secondary Endpoint(s) | 9 |
| | 1.2.4 | Safety Endpoints | 10 |
| | 1.2.5 | Safety Endpoints Other Endpoints .5.1 PK Endpoint imand(s) Y DESIGN | 11 |
| | 1.2 | .5.1 PK Endpoint | 11 |
| 1 | 3 Est | imand(s) | 11 |
| 2.0 | STUD | Y DESIGN | 11 |
| 3.0 | STATI | STICAL HYPOTHESES AND DECISION RULES | 13 |
| 4.0 | | LE-SIZE DETERMINATION | |
| 5.0 | ANAL | YSIS SETS | 13 |
| 5. | 1 All | Subjects Who Signed the Informed Consent Form | 13 |
| 5.2 | 2 All | Subjects Who Did Not Enter the Treatment Period | 13 |
| 5 | 3 Saf | Fety Analysis Set | 14 |
| 5.4 | 4 Inte | ention-to-treat set (ITT) | 14 |
| 5.: | 5 Per | Protocol Analysis Set (PPS) | 14 |
| 6.0 | STATI | STICAL ANALYSIS | 14 |
| 6. | _0 | neral Considerations | |
| 6.2 | 2 An | alysis Approach | 16 |
| Ç, | 6.2.1 | Analysis Cohort | 16 |
| , 0) | 6.2.2 | Analysis Approach for Continuous Efficacy Endpoints | 17 |
| (5) | 6.2.3 | Analysis Approach for Binary Efficacy Endpoints | 17 |
| | 6.2.4 | Analysis Approach for Time-to-Event Efficacy Endpoints | 17 |
| 6 | 3 Dis | sposition of Subjects | 17 |
| | 6.3.1 | Study Information | 17 |
| | 632 | Screen Failures | 18 |

| | 6.3 | .3 | Subj | ect Eligibility | 18 |
|---|---|---|---|---|---|
| | 6.3 | .4 | Num | ber of Subjects Who Entered the Treatment Period by Site | 18 |
| | 6.3 | .5 | Disp | osition of Subjects | 19 |
| | 6.3 | .6 | Proto | ocol Deviations and Analysis Sets | . 19 |
| | | 6.3.6 | 5.1 | Significant Protocol Deviations | 19 |
| | | 6.3.6 | 5.2 | Analysis Sets | 20 |
| 6.4 | | Dem | ograp | phic and Other Baseline Characteristics | 20 |
| | 6.4 | .1 | Dem | Analysis Sets | 20 |
| | 6.4 | 2 | Med | ical History and Concurrent Medical Conditions | 23 |
| 6.5 | | Med | icatio | on History and Concomitant Medications | 23 |
| 6.6 | | Exte | nt of | Exposure and Compliance | 24 |
| 6.7 | | Effic | acy A | Analysis | 24 |
| | 6.7 | '.1 | Prim | ary Endpoint Analysis | 24 |
| | | 6.7.1 | .1 | Primary Analysis | 24 |
| | | 6.7.1 | .2 | Exposure and Compliance Analysis ary Endpoint Analysis Primary Analysis Sensitivity Analysis Supplementary Analyses andary Endpoints Analysis Manalysis | 24 |
| | | 6.7.1 | 3 | Supplementary Analyses | 25 |
| | 6.7 | .2 | Seco | ondary Endpoints Analysis | 25 |
| | | 0.7.2 | I | Key Secondary Endpoints | 25 |
| | | 6.7.2 | | Sensitivity Analysis. | |
| | | 6.7.2 | 2.3 | Secondary Endpoints | 26 |
| | | | 4.0 | | |
| | 6.7 | | _ | group Analysis | |
| 6.8 | | - (_) | | alysis | |
| | 6.8 | | | erse Events | |
| ٠, | 10 | 6.8.1 | | Overview of Treatment-Emergent Adverse Events | |
| 0, | | 6.8.1 | | Displays of Treatment-Emergent Adverse events | |
| 4 | | 6.8.1 | | Displays of Pretreatment Events | |
| | 6.8 | | | ical Laboratory Evaluations | |
| | | 6.8.2 | | Laboratory Tests other than Urinalysis | |
| | | 6.8.2 | | Urinalysis | |
| | 6.8 | .3 | Vital | Signs, Weight and Height | 33 |

| | 6.8.4 | ECGs | 34 |
|---|---|---|---|
| | 6.8.5 | Displays of Treatment-Emergent Adverse Events (Japanese) | |
| 6.9 | Pha | rmacokinetic, Pharmacodynamic, and Biomarker Analyses | |
| | 6.9.1 | Pharmacokinetic Analysis | 35 |
| | 6.9. | Pharmacokinetic Analysis | 35 |
| 6.10 | 0 Oth | er Analyses | 35 |
| | 6.10.1 | Analyses for Overall Supplemental Cohort. Analyses for All Cohorts Combined ENCES | 35 |
| | 6.10.2 | Analyses for All Cohorts Combined | 35 |
| 7.0 | REFER | ENCES | 36 |
| 8.0 | CHANG | GES TO PROTOCOL PLANNED ANALYSES | 36 |
| 9.0 | APPEN | DIX | 36 |
| 9.1 | Cha | nges From the Previous Version of the SAP | 36 |
| 9.2 | Data | Handling Conventions Definition of Study Days Definition of Study Visit Windows | 49 |
| | 9.2.1 | Definition of Study Days | 49 |
| | 9.2.2 | Definition of Study Visit Windows | 50 |
| | 9.2. | 2.1 Endpoints other than ItchRO Scores and PK Samples | 50 |
| | 9.2. | 2.2 PK Samples | 53 |
| | 9.2. | 2.3 Average ItchRO Scores | 54 |
| | 9.2.3 | Partial Date Conventions. | |
| 9.3 | Der | vation of Endpoints | 56 |
| | 9.3.1 | Primary Efficacy Endpoints | 56 |
| | 9.3.2 | Average ItchRO Scores | 56 |
| | 9.3.3 | Responder Endpoints | 57 |
| | 9.3.5 | Z-scores | 58 |
| | 9.3.6 | Lists of Laboratory Tests | |
| | 9.3.7 | Table for AECI | |
| | 9.3.8 | Significance Level and Confidence Coefficient | |
| 9.4 | Ana | lysis Software | 59 |
| O | | | |
| LIST ( | OF IN-T | TEXT TABLES | |
| Table 9 | ).1 | Visit Window of sBA, sBA subspecies, C4, Serum Storage Sample | 50 |
| Table 9 | | Visit Window of Vital Signs, Weight and Height, | |
| | | | 51 |
| Table 9 | 0.3 | Urinalysis, Cholestasis Biomarkers (FGF19) | 51 |

| | 2 Pag<br>alysis Plan 2.0 10 |
|---|---|
| Table 9.4 | Lipid Panel, Lipid Soluble Vitamins |
| Table 9.5 | CBC, Coagulation, Chemistry Panel |
| Table 9.6 | Visit Window of ECGs, AFP |
| Table 9.8 | Visit Window of PK |
| Table 9.9 | Visit Window of Average ItchRO Score |
| LIST OF IN | Visit Window of Average ItchRO Score N-TEXT FIGURES Schematic Study Design |
| LIST OF IT | Schematic Study Design |
| | ial use only |
| | ,()* |
| | non-commerc. |
| | 28. For non-commerco |
| 1 of the | da. For non-commerco |
| of the state of th | ada. For non-corninero |
| is of the | da. For non-commerce |
| X) STAPE | ada. For non-commerc. |
| is of the | Lipid Panel, Lipid Soluble Vitamins CBC, Coagulation, Chemistry Panel Visit Window of ECGs, AFP |

Page 7 of 59

10Nov2023

## **ABBREVIATIONS**

AE adverse event

**AECI** adverse event of clinical interest

**AFP** alpha-fetoprotein ALP alkaline phosphatase alanine aminotransferase ALT ANCOVA analysis of covariance APRI AST to platelet ratio index

aPTT activated partial thromboplastin time

AST aspartate aminotransferase 7αC4 7α-hydroxy-4-cholesten-3-one

body mass index BMI BUN blood urea nitrogen CBC complete blood count confidence interval CI

**ECG** Electrocardiogram

fibroblast growth factor 190 FGF-19

fibrosis-4 FIB-4

gamma-glutamyl transferase GGT **HCC** hepatocellular carcinoma

high density lipoprotein-cholesterol HDL-C

health-related quality of life **HRQoL** 

ItchRO Observer ItchRO(Obs) ItchRO Patient ItchRO(Pt) ITT intention-to-treat set

KM Kaplan-Meier

low density lipoprotein-cholesterol LDL-C

lower limit of normal

last observation carried forward LOCF

XIS means least square means LSV lipid soluble vitamin

**MCH** mean corpuscular hemoglobin

mean corpuscular hemoglobin concentration **MCHC** 

**MCV** mean corpuscular volume MedDRA Medical Dictionary for Regulatory Activities

**MITT** modified intention-to-treat set **PEBD** partial external biliary diversion

progressive familial intrahepatic cholestasis **PFIC** 

PK pharmacokinetic

PPS per-protocol analysis set PRO patient-reported outcomes

PT preferred term 25th percentile Q1 75th percentile Q3

QT interval corrected using Bazett's formula **QTcB** QTcF QT interval corrected using Fridericia's formula only and suf

QOL quality-of-life

RBP retinol binding protein serious adverse event SAE SAP statistical analysis plan

sBA

serum bile acid serum glutamic-oxaloacetic transaminase **SGOT** serum glutamic-pyruvic transaminase **SGPT** 

SOC system organ class

TEAE treatment-emergent adverse event

triglycerides TG

WBC
WHODrug total serum bilirubin upper limit of normal white blood cell

World Health Organization Drug Dictionary

### 1.0 **OBJECTIVES, ENDPOINTS AND ESTIMANDS**

### 1.1 **Objectives**

### 1.1.1 **Primary Objective**

- To evaluate the efficacy of TAK-625 in the primary cohort.
- To evaluate the safety of TAK-625 in subjects with PFIC.

### 1.1.2 **Secondary Objective(s)**

- To evaluate the efficacy of TAK-625 in subjects with PFIC.
- To evaluate the PK of TAK-625 in subjects with PFIC.

### 1.1.3 Additional Objective(s)

applicable Terms of Use To evaluate primary, secondary, and exploratory endpoints in the supplemental cohort

### 1.2 **Endpoints**

### 1.2.1 **Primary Endpoint(s)**

Change in the average morning ItchRO (Obs) severity score between baseline and average of Week 15 through Week 26.

### 1.2.2 Secondary Endpoint(s)

### 1.2.2.1 Key Secondary Endpoints(s)

- Change in the average morning ItchRO (Obs) frequency score between baseline and average of Week 15 through Week 26.
- Change in total sBA between baseline and Week 26

### 1.2.2.2 Secondary Endpoint(s)

- Proportion of subjects who experience an sBA control (defined as a reduction to <102 $\mu$ mol/L, or a reduction of >75%, or normalization) from baseline through Week 26.
- Change in the ItchRO (Obs) weekly average severity (based on daily maximum of morning and evening severity scores) between baseline and average of Week 15 through Week 26.



# 1.2.4 Safety Endpoints

• Incidence of AEs including SAEs, related to study drug, leading to study drug discontinuation, and AEs of clinical interest (AECIs).

AECIs include the following:

- LSV deficiency events.
- Liver parameter disruption.
- ns of Use Change from baseline in clinical laboratory values (hematology, chemistry, urinalysis, and others), physical examination findings (including body weight, height, and body mass index [BMI]), vital signs, and electrocardiogram (ECG) parameters

### 1.2.5 **Other Endpoints**

### 1.2.5.1 PK Endpoint

- Plasma levels of TAK-625 at predose and approximately 2.5 hours after the morning dose at Week 10.
- Plasma levels of TAK-625 at predose (optional) and approximately 30 minutes after morning dose at Week 14 (or any visit up to Week 26).

### 1.3 Estimand(s)

Not Applicable.

### 2.0 STUDY DESIGN

This is a phase 3, multicenter, open-label, uncontrolled study to evaluate the efficacy and safety of TAK-625 in the treatment of Japanese subjects with PFIC. Study Population:

The study population is defined as Japanese patients with PFIC who are 1 year of age or older". Subjects diagnosed with PFIC2 due to ABCB11 mutation that predicts residual BSEP function (nt-PFIC2) will be enrolled in the primary cohort. Subjects with other PFIC subtypes (eg, t-PFIC2, PFIC1/3/4, or other PFIC mutation variants) or postsurgical subjects (eg, internal or external biliary diversion surgery) will be enrolled in the supplemental cohort. (Subjects diagnosed with PFIC2 due to ABCB11 mutation that predicts complete absence of BSEP function [t-PFIC2] are excluded from the primary cohort and can be enrolled only in the supplemental cohort. PFIC subtypes should be determined by a genotyping [refer to Protocol Section 7.11).

Study Period (Screening, Treatment [Dose Escalation, Stable Dosing, and Follow-Up Dosing], and Safety Follow-Up Period):

This study consists of the screening period (up to 6 weeks prior to the study administration), 💞 4 week dose escalation period (doses up to 600 ug/kg, BID, as tolerated), 44-week stable dosing period, and follow-up dosing period (until TAK-625 is approved or available in Japan commercially, or if the subject withdraws from the study, or if the investigator determines the subject's discontinuation, or if the sponsor stops the program or development in this indication).

1. Screening Period (up to 6 Weeks prior to the Study Administration):

In the screening period, for subjects who do not have documentation of mutation related with PFIC, a blood sample will be obtained for genotyping. Subjects diagnosed with PFIC2 (nt-PFIC2) will be enrolled in the primary cohort and those with other types of PFIC will be enrolled in the supplemental cohort. The electronic Diary (eDiary) for assessing pruritus with the Itch Reported Outcome (ItchRO) instrument will be dispensed and subjects and caregivers will undergo training during the screening visit.

# 2. Dose Escalation Period (4 weeks [up to 6 weeks]: Week 0 to 4 [6]):

In the dose escalation period, at the baseline visit (Week 0/Visit 2), subjects will be assessed to confirm continued study eligibility and undergo a physical examination including body weight, height, BMI, and vital signs, and have urine and blood samples taken for hematology, chemistry, fasting lipid panel, baseline levels of sBA and other cholestasis biochemical markers. Compliance with ItchRO will be assessed. Study drug will be supplied at each visit (Week 0/Visit 2, Week 2/Visit 3, and Week 4/Visit 4). The subject contacts (phone calls) will be conducted at Weeks 1 and 3. The dose is increased weekly, 150 µg/kg, 300 µg/kg, 450 µg/kg, and 600 µg/kg, BID.

Dose escalation should occur in the absence of major safety (eg, liver parameters and LSV deficiency) or tolerability concerns (eg, GI-related TEAEs) related or possibly related to study drug. Subjects with such safety concerns can be down-titrated to a lower, previously tolerated dose level for 1 week before continuing dose escalation. The minimum dose to continue in the study will be  $150 \, \mu \text{g/kg}$ , BID; subjects who cannot tolerate this dose will be discontinued from the study. The dose escalation period is allowed to be extended up to 6 weeks depending on the safety or tolerability concerns (refer to Protocol Section 8.1.3).

# 3. Stable Dosing Period (44 weeks: Week 5 to 48):

After the dose escalation period, each subject will continue dosing with study drug at the Week 4 or Week 6 dose level (the maximum tolerated dose [MTD] level) in the stable dosing period. Subjects will return to the study site at Weeks 6, 10, 14, 18, 22, 26, 28, 32, 36, 40, 44, and 48 and undergo physical examinations. Subject contacts (phone calls) will be conducted as appropriate throughout the stable dosing period. Subjects and caregivers will continue twice daily completion of their ItchRO throughout the period.

# 4. Follow-up Dosing Period (after Week 48):

Additionally, in the follow-up dosing period, each subject will continue dosing with study drug. The safety evaluation will be performed in all the subjects every 12 weeks from Week 48 visit until TAK-625 is approved or available in Japan commercially, or if the subject withdraws from the study, or if the investigator determines the subject's discontinuation, or if the sponsor stops the program or development in this indication. Bile acids and ItchRO will be measured to evaluate the long-term effectiveness of TAK-625. For subjects discontinuing early, safety follow-up will be conducted.

# 5. Safety Follow-up (after Final Visit/ET):

Subjects/caregivers will have a final safety follow-up subject contact (phone call) 7 days after the final study visit or ET visit (except for screen failure).

A schematic of the study design is included as Figure 2.a. A schedule of assessments is listed in Protocol Appendix A.

Figure 2.a Schematic Study Design



ID=twice daily, SCR=screening, W=week, wks=weeks

# 3.0 STATISTICAL HYPOTHESES AND DECISION RULES

Not Applicable.

# 4.0 SAMPLE-SIZE DETERMINATION

PFIC is a rare disease. The targeted sample size of the primary cohort is approximately 3 subjects, and that of the supplemental cohort is approximately 6 subjects, based on enrollment feasibility of this population in Japan, rather than power calculation.

# 5.0 ANALYSIS SETS

# 5.1 All Subjects Who Signed the Informed Consent Form

All subjects who signed the informed consent form.

# 5.2 All Subjects Who Did Not Enter the Treatment Period

All subjects who did not enter the treatment period.

### 5.3 Safety Analysis Set

All subjects who received at least one dose of study drug.

### 5.4 **Intention-to-treat set (ITT)**

All subjects who received at least one dose of study drug.

### 5.5 **Per-Protocol Analysis Set (PPS)**

ble Lekins of Use All ITT subjects who did not have any of the following major protocol deviations and whose primary endpoint was evaluable primary endpoint was evaluable.

- Subjects who did not meet inclusion criteria #3, 4, 5, 6.
- Subjects who met exclusion criteria #1,2, 3, 4, 5, 6, 7, 9, 15, 16, 17, 19

### STATISTICAL ANALYSIS 6.0

Statistical analyses will be performed using all subjects' data up to Week 26 (i.e., up to Day 197) after the data are locked. PK analysis will be performed using all subjects' data up to Week 10 after the data are locked.

### 6.1 **General Considerations**

The following definitions and calculation formulas will be used.

- **Treatment-emergent adverse event (TEAE)**: An adverse event whose date of onset occurs on or after the start of study drug, TEAEs whose date of onset occurred on or before Week 26 visit (i.e. the latest visit by Day 197), will be summarized.
- Pretreatment event (PTE): Any untoward medical occurrence in a clinical investigation subject who has signed informed consent to participate in a study but prior to administration of study drug.
- Concomitant medication: Concomitant medications whose start date occurred on or before Week 26 visit (i.e. the latest visit by Day 197), will be summarized.
- Descriptive statistics for endpoints other than PK: Number of subjects, mean, standard deviation, standard error, maximum, minimum, and quartiles (Q1, median, and Q3).
- Descriptive statistics for PK: Number of subjects, mean, standard deviation, maximum, median, minimum, coefficient of variation, and geometric mean.
  - Duration of exposure to study drug (days): {Date of last dose of study drug or Week 26 visit (i.e. the latest visit by Day 197) which comes faster - date of first dose of study drug} +
- Duration of study after baseline (days): {Date of last visit/contact or Week 26 visit (i.e. the latest visit by Day 197) which comes faster - date of first dose of study drug} + 1.

- Study drug compliance (%): Number of study drugs taken / (duration of exposure to study drug \* 2) \* 100 (rounded to 1 decimal place).
- **Dose Level (μg/kg)**: Strength of study drug taken (mg) / (last available body weight (kg) prior to or on the day of study drug taken) \* 1000.
- **Dose Level Categories for PK (µg/kg)**: Categorize by following below calculation rule. If Min <= dose level < 225 µg/kg, then dose level category = 150 µg/kg; if 225 µg/kg <= dose level < 375 µg/kg, then dose level > category = 300 µg/kg; if 375 µg/kg <= dose level < 525 µg/kg, then dose level category = 450 µg/kg; if 525 µg/kg <= dose level <= Max, then dose level category = 600 µg/kg.
- Total Drug Exposure (μg/kg): Sum of {number of study drugs taken \* dose level received (μg/kg)}.
- **Average Daily Dose (μg/kg/day)**: Total Drug Exposure (μg/kg) / Duration of exposure to study drug (days).
- ItchRO (Obs/Pt) Daily Maximum of Morning and Evening Scores: Maximum of morning and evening severity scores for each day. The morning and evening severity scores of the same day should be used for the calculation. Both the morning and evening ItchRO reports have a minimum score of 0 and a maximum score of 4, with 4 representing more severe (Item 1) itching.
- **Time to liver-associated events**: PEBD surgery, listing for liver transplantation, liver decompensation [hepatic encephalopathy, variceal bleeding, ascites, and spontaneous bacterial peritonitis] events, hepatocellular carcinoma (HCC), death, and other.
- Estimated Total Lipids (mg/dL): Cholesterol (mg/dL) + Triglycerides (mg/dL)
- Ratio of Alpha-tocopherol to Estimated Total Lipids (mg/g): 1000 \* Alpha-tocopherol (mg/dL) / Estimated Total Lipids (mg/dL). For Alpha-tocopherol concentrations reported as below the minimum quantitation limit, half of the minimum quantitation limit is used in the calculation.
- Corrected Sodium (mEq/L): sodium (mEq/L) + (0.002 \* Triglycerides (mg/dL)).
- FIB-4: (Age (years) \* AST (U/L)) / (platelet count  $(10^9/L)$  \* sqrt(ALT(U/L)))
  - Age (years) is years at sample collection visit.
- APRI:  $100 * (AST (U/L) / AST ULN(U/L)) / (platelet count (10^9/L))$ 
  - ULN is upper limit normal
- **Significant Protocol Deviation**: Deviation defined in the PDMP as "Important PD" whose Severity Classifications is "major" or "critical".
- Time since original diagnosis of PFIC (months): (date of first dose date of original diagnosis of PFIC + 1) / 30.4375.

When reporting derived values or parameters, following presenting rules will be applied.

- For sBA, ItchRO: For rules on rounding and decimal presentation of these statistics, along with the rules for presenting certain derived values see below.
  - For measures of median and mean, use 3 decimal places.
  - For measures of standard deviation, standard error of the mean and CI, use 4 decimal places.
  - For measures of minimum and maximum values as well as observed value (for Listing), use 2 decimal places.
  - >=5 is rounded up away from zero, whereas <5 is rounded down toward zero, to account for rounding of negative numbers.
  - For p-values use 3 decimal places.
  - $\triangleright$  Presentation of p-values display p-values that would round to 0.000 as <0.001.
- Other than sBA, and ItchRO: For rules on rounding and decimal presentation of these statistics, along with the rules for presenting certain derived values see below.
  - For measures of median and mean, use 1 decimal place beyond those used for the measurement.
  - For measures of standard deviation, standard error of the mean and CI, use 2 decimal places beyond those used for the measurement.
  - For measures of minimum and maximum values, use the same number of decimal places as those used for the measurement.
  - >=5 is rounded up away from zero, whereas <5 is rounded down toward zero, to account for rounding of negative numbers.
  - For p-values use 3 decimal places.
  - $\triangleright$  Presentation of p-values display p-values that would round to 0.000 as <0.001.
  - > BMI should be rounded to 1 decimal place for reporting.
  - > Derived questionnaire scores, and other similar efficacy parameters recorded as integers, should be rounded to 1 decimal place for reporting.
  - Averaged lab results (e.g. Diastolic/Systolic Blood Pressure and Pulse [when taken in triplicate]) should be rounded to 1 decimal place for reporting.

# Analysis Approach

# 6.2.1 Analysis Cohort

Analyses described in section  $6.3 \sim 6.9$  will be performed for primary cohort.

### 6.2.2 **Analysis Approach for Continuous Efficacy Endpoints**

For efficacy endpoints, all continuous endpoints in this trial will use the analysis method below unless stated otherwise in the section specific to an endpoint.

Descriptive statistics and two-sided 95% confidence interval of mean will be provided for observed values (baseline and post-baseline visits) and changes from baseline (each postbaseline visit - baseline). For endpoint with multiple visits, these will be provided by visit.

### 6.2.3 **Analysis Approach for Binary Efficacy Endpoints**

For efficacy endpoints, all binary endpoints in this trial will use the analysis method below unless stated otherwise in the section specific to an endpoint.

Frequency distribution will be provided by visit, with proportion and the two-sided 95% confidence interval. For endpoint with multiple visits, these will be provided by visit.

### 6.2.4 Analysis Approach for Time-to-Event Efficacy Endpoints

For efficacy endpoints, all time-to-event endpoints in this study will use the analysis method below unless stated otherwise in the section specific to an endpoint.

The event-free survival rate and the two-sided 95% confidence intervals will be provided using the Kaplan-Meier method. The event-free survival rate will also be plotted. Time to event will be defined as the date of first dose of study drug to the event which comes fastest. For subjects without an event, time to event will be defined as the date of first dose of study drug to the censoring date, which is the date of the last study visit/contact.

### **Disposition of Subjects** 6.3

# Study Information 6.3.1

All Subjects Who Signed the Informed Consent Form Analysis Set:

Analysis Endpoint(s) Date First Subject Signed Informed Consent Form

Date of Last Subject's Last Visit/Contact

MedDRA Dictionary Version

WHO Drug Dictionary Version

SAS Version Used for Creating the Datasets

Analytical Method(s): (1) Study Information

Study information shown in the analysis endpoints section will be

provided.

### 6.3.2 **Screen Failures**

Analysis Set: All Subjects Who Did Not Enter the Treatment Period

Analysis Endpoint(s): Age (years)

> Gender [Male, Female]

Analytical Method(s): (1) Screen Failures

Frequency distributions for categorical endpoints and descriptive

statistics for continuous endpoints will be provided.

### 6.3.3 **Subject Eligibility**

All Subjects Who Signed the Informed Consent Form Analysis Set:

[Eligible for Entrance into the Analysis Endpoint(s): **Eligibility Status** 

> Treatment Period, Not Eligible for Entrance into the Treatment Period]

Primary Reason for Subject

Not Being Eligible

JAE, Screen Failure (Did not meet inclusion criteria or did meet exclusion criteria), Protocol

Deviation, Lost to Follow-up, Pregnancy, Withdrawal by Subject, Study Terminated by Sponsor, Other]

(1) Eligibility for Entrance into the Treatment Period Analytical Method(s):

Frequency distributions will be provided. When calculating

percentages for the primary reasons for subject not being eligible, the total number of ineligible subjects will be used as the denominator.

### Number of Subjects Who Entered the Treatment Period by Site 6.3.4

Analysis Set: ITT

Analysis Endpoint(s): Status of Entrance into the [Entered]

Treatment Period

Site [Site numbers will be used as

categories]

Analytical Method(s): (1) Number of Subjects Enrolled by Site

Frequency distribution will be provided for each stratum.

### 6.3.5 **Disposition of Subjects**

ITT Analysis Set:

Analysis Endpoint(s): Study Drug Completion

Status

[Ongoing, Completed Study Drug,

Prematurely Discontinued Study

Drug]

Reason for Discontinuation

of Study Drug

[AE, Protocol Deviation, Lost to Follow-up, Withdrawal by Subject, Study Terminated by Sponsor,

Pregnancy, Lack of Efficacy, Other]

Completion Status of All

Planned Study Visits

[Ongoing, Completed Study, Prematurely Discontinued Study]

Reason for Discontinuation

of Study

[AE, Protocol Deviation, Lost to Follow-up, Withdrawal by Subject, Study Terminated by Sponsor,

Pregnancy, Lack of Efficacy, Other]

(1) Disposition of Subjects Analytical Method(s):

> Frequency distributions will be provided. When calculating percentages for the reasons for discontinuation, the total number of

subjects who prematurely discontinued will be used as the

denominator.

### 6.3.6 **Protocol Deviations and Analysis Sets**

Significant Protocol Deviations 6.3.6.1

Analysis Set:

Analysis Endpoint(s) Significant Protocol Deviation [Informed Consent and Process,

Inclusion Criteria, Exclusion Criteria, Concomitant Medication, Laboratory Assessment, Study Procedures (not safety and efficacy related), Safety, Visit Schedule, IP conditions, IP preparation, IP administration, Subject IP Compliance, Efficacy,

Subject Discontinuation,

Administrative, Patient Reported Outcomes, PK/PD, Other Criteria]

Property of Takeda. Analytical Method(s): (1) Protocol Deviations

re of Use Frequency distribution will be provided for each deviation category. A subject who has several deviations will be counted once in each appropriate category. A subject who has several deviations that can be classified into the same category will be counted only once.

### 6.3.6.2 Analysis Sets

Analysis Set: ITT

Analysis Endpoint(s):

[Categories are based on the definitions in Handling of Subjects

Section 5.0]

**Analysis Sets** 

ITT [Included]

**PPS** [Included]

[Included] Safety Analysis Set

(1) Subjects Excluded from Analysis Sets Analytical Method(s):

(2) Analysis Sets

Frequency distributions will be provided. For (1), a subject who has several reasons for exclusion will be counted once in each appropriate category. A subject who has several reasons for exclusion that can be classified into the same category will be counted only once.

### 6.4 **Demographic and Other Baseline Characteristics**

### **Demographic and Baseline Characteristics** 6.4.1

Analysis Set:

Property of Lakedai. Analysis Endpoint(s): [Min<= - < 9, 9<= - <= 18, 18< -Age (years)

 $\leq Max$ 

 $[Min \le - <7, 7 \le - \le Max]$ 

Gender [Male, Female]

Height (cm)

Weight (kg)

BMI (kg/m2)

Height z-score

Weight z-score

and subject to the applicable Terms of Use BMI z-score Time Since Original Diagnosis of PFIC, in Months Used Anything to Treat Itch in the Past Type of Therapy Used to Treat Itch in the Past (multiple count) **Topical** Oral Other Specific Therapy Used to Treat Itch in the Past Topical Corticosteroids Topical Calcineurin **Inhibitors Topical Antihistamines** Menthol Capsaicin

Property of Takeda. For non's **Local Anesthetics** Androgens Anticholestatic Agents Anticonvulsants Antidepressants Antihistamines Anti-Oxidants **Binding Resins** 

Salicylic acid

Colchicine

Cannabinoid Agonist

**Enzyme Inducers** 

**Immunosuppressants** 

**Opiate Antagonists** 

Serotonin Antagonists

Ursodeoxycholic Acid

**IBAT Inhibitors** 

Surgical Interruption of the **Enterohepatic Circulation** 

Phototherapy

Hemofiltration

Plasmapheresis

Nasal Biliary Drainage

Other

ItchRO(Obs) 4-week

Morning

[PFIC1, PFIC2, PFIC3, PFIC4,

PFIC5, PFIC6]

(1) Demographics and Baseline Characteristics

erity (Item

LhRO(Obs) 4-week

Morning

Average Frequency (Item 3)

Score

SBA (LC MS)

PFIC Subtype

Analytical Method(s): (1) Frequency distributions for categorical endpoints and descriptive statistics for continuous endpoints will be provided. PFIC subtype will be provided in Section 6.10.1 and 6.10.2 only.

### 6.4.2 **Medical History and Concurrent Medical Conditions**

ITT Analysis Set:

Analysis Endpoint(s): Medical History

Concurrent Medical Conditions

ierms of Use (1) Medical History by System Organ Class and Preferred Term Analytical Method(s):

> (2) Concurrent Medical Conditions by System Organ Class and Preferred Term

Frequency distributions will be provided. MedDRA dictionary will be used for coding. Summaries will be provided using SOC and PT, where SOC will be sorted alphabetically and PT will be sorted in decreasing frequency.

A subject with multiple occurrences of medical history or concurrent medical condition within a SOC will be counted only once in that SOC. A subject with multiple occurrences of medical history or concurrent medical condition within a PT will be counted only once in that PT.

### **Medication History and Concomitant Medications** 6.5

(1) Medication History by Anatomical Therapeutic Chemical Level 2

Ongoing at Baseline as well as Those That Started After Baseline

Medication History by Anatomical Therapeutic Chemical Land Preferred Medication Name

(2) Concomitant Medications That Started and Stopped Prior to Baseline by Anatomical Therapeutic Chemical Level 2 and Preferred Medication Name

(3) Concomitant Medications That Started Prior to Congoing at Baseline as well as Those The by Anatomical Therapeutic Chemical Chemical Therapeutic Chemical Level 2 and Preferred Medication Name

Frequency distributed the Started Prior to Chemical Level 2 and Preferred Medication Name

Frequency distributed the Started Pri Frequency distributions will be provided. WHO Drug dictionary will be used for coding. Summaries will be provided using anatomical subject who has been administered several medications with the same preferred medication names will be counted only once for that preferred medication names. For anatomical therapeutic chemical level 2, same manners in counting frequency.

# **Extent of Exposure and Compliance**

Analysis Set: ITT

Analysis Endpoint(s): Duration of Exposure to  $[0 \le - \le 28, 29 \le - \le Max]$ 

Study Drug (days)

Study Drug Compliance (%) [Min<= - < 80, 80 <= - <= 100, 100<

<=Max

Total Drug Exposure (µg/kg)

Average Daily Dose

 $(\mu g/kg/day)$ 

Analytical Method(s): (1) Study Drug Exposure, Compliance, Total Drug Exposure and

Average Daily Dose

Frequency distributions for categorical endpoints and descriptive

statistics for continuous endpoints will be provided.

is

oint Analysis

ysis

ITT

# 6.7 Efficacy Analysis

# 6.7.1 Primary Endpoint Analysis

# 6.7.1.1 Primary Analysis

Analysis Set: ITT

Analysis Endpoint(s): Change in the average morning ItchRO (Obs) severity score between

baseline and average of Week 15 through Week 26

Analytical Method(s): See Section 6.2.2.

# 6.7.1.2 Sensitivity Analysis

Analysis Set: PPS

Analysis Endpoint(s): Change in the average morning ItchRO (Obs) severity score between

baseline and average of Week 15 through Week 26

Analytical Method(s): See Section 6.2.2. For supportive analysis the same analysis as the

primary analysis will be performed using the PPS to confirm

robustness of the results.

# 6.7.1.3 Supplementary Analyses

Analysis Set: ITT

Analysis Endpoint(s): Change in the average morning ItchRO (Obs) severity score between

baseline and average of Week 15 through Week 26

Analytical Method(s): If possible, the endpoint will be analyzed using a MMRM model. The

repeated measures include post-baseline visits (i.e., Week 6, 10, 14, 18, 22, and 26), with change from baseline in the 6- or 4-week average morning ItchRO(Obs) severity score as the response. The MMRM will also include visit, baseline and baseline-by-visit interaction as fixed effects. LS means and the two-sided 95%

confidence intervals will be provided using the contrast across the last 12 weeks of the study (i.e., Weeks 18, 22, and 26 combined). In other words, the analytical solution from the MMRM is an equally weighted average of the 3 individual visit-specific estimates over the time

period of interest (i.e., Weeks 18, 22, and 26).

The unstructured variance/covariance matrix will be used to model the variances and covariances. However, if the numerical algorithm for estimation of the mixed model fails to converge, the alternative

variance/covariance matrix structures will be used (e.g.,

heterogeneous autoregressive of order 1). The Kenward-Roger approximation will be used to estimate denominator degrees of

freedom.

# 6.7.2 Secondary Endpoints Analysis

# 6.7.2.1 Key Secondary Endpoints

Analysis Set:

\_YTT

Analysis Endpoint(s)

- Change in the average morning ItchRO (Obs) frequency score between baseline and average of Week 15 through Week 26
- Change in total sBA between baseline and Week 26

Analytical Method(s):

See Section 6.2.2.

### 6.7.2.2 Sensitivity Analysis

Analysis Set:

**PPS** 

Analysis Endpoint(s):

Change in the average morning ItchRO (Obs) frequency score between baseline and average of Week 15 through Week 26

Change in total sBA between baseline and Week 26

Analytical Method(s):

See Section 6.2.2. For supportive analysis the same analysis as the primary analysis will be performed using the PPS to confirm to the abb robustness of the results.

### 6.7.2.3 Secondary Endpoints

Analysis Set:

ITT

Analysis Endpoint(s):

Analytical Method(s):

Proportion of subjects who experience an sBA control

Change in the ItchRO (Obs) weekly average severity (based on daily maximum of morning and evening severity scores) between baseline and average of Week 15 through Week 26

See Section  $6.2.2 \sim 6.2.3$ 





# 6.7.4 Subgroup Analysis

Analysis Set:

ITT

Analysis Endpoint(s):

- Change in the average morning ItchRO (Obs) severity score between baseline and average of Week 15 through Week 26
- Change in the average morning ItchRO (Obs) frequency score between baseline and average of Week 15 through Week 26
- Change in total sBA between baseline and Week 26

Subgroup(s):

Age

 $[Min \le - <7, 7 \le - \le Max]$ 

Gender

[Male, Female]

applicable Terms of Use Descriptive statistics will be provided for above each subgroup. Analytical Method(s):

### 6.8 **Safety Analysis**

### 6.8.1 **Adverse Events**

6.8.1.1 Overview of Treatment-Emergent Adverse Events

Analysis Set: Safety Analysis Set

Analysis Endpoint(s): **TEAE** 

[Related, Not Related] Categories: Relationship to Study Drug

> [Mild, Moderate, Severe] Intensity

The following summaries will be provided. Analytical Method(s):

(1) Overview of Treatment-Emergent Adverse Events

- 1) All Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
- Relationship of Treatment-Emergent Adverse Events to study drug (number of events, number and percentage of subjects)
- 3) Intensity of Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
- Treatment-Emergent Adverse Events leading to study drug discontinuation (number of events, number and percentage of subjects)
- Serious Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
- 6) Relationship of serious Treatment-Emergent Adverse Events to study drug (number of events, number and percentage of subjects)
- 7) Serious Treatment-Emergent Adverse Events leading to study drug discontinuation (number of events, number and percentage of subjects)
- Treatment-Emergent Adverse Events resulting in death (number of events, number and percentage of subjects)

Property of Takeda. For non-com
TEAEs will be counted according to the rules below.

#### Number of subjects

- Summaries for 2) and 6)
   A subject with occurrences of TEAE in both categories (i.e., Related and Not Related) will be counted once in the Related category.
- Summary for 3)
   A subject with multiple occurrences of TEAE will be counted once for the TEAE with the maximum intensity.
- Summaries other than 2), 3), and 6)
  A subject with multiple occurrences of TEAE will be counted only once.

#### Number of events

For each summary, the total number of events will be calculated.

### 6.8.1.2 Displays of Treatment-Emergent Adverse events

Analysis Set: Safety Analysis Set

Analysis Endpoint(s): TEAE

Property of Takeda. For

Categories: Intensity [Mild, Moderate, Severe]

Time of Onset (day) [1-28, 29 - Max]

Analytical Method(s): The following summaries will be provided using frequency

distribution.

TEAEs will be coded using the MedDRA and will be summarized using SOC and PT.

SOC will be sorted alphabetically and PT will be sorted in decreasing frequency for tables provided by SOC and PT. SOC and PT will be sorted in decreasing frequency for tables provided by System Organ Class only or PT only.

- (1) Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (2) Treatment-Emergent Adverse Events by System Organ Class
- (3) Treatment-Emergent Adverse Events by Preferred Term
- (4) Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term

- (5) Intensity of Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (6) Intensity of Drug-Related Treatment-Emergent Adverse Events by System Organ Class, and Preferred Term
- (7) Treatment-Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term
- (8) Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (9) Treatment-Emergent Adverse Events by System Organ Class and Preferred Term Over Time
- (10) Treatment-Emergent Adverse Events of Clinical Interest by System Organ Class and Preferred Term
- (11) Drug-Related Treatment-Emergent Adverse Events of Clinical Interest by System Organ Class and Preferred Term

The frequency distribution will be provided according to the rules below.

### Number of subjects

- Summary tables other than (5), (6) and (9) A subject with multiple occurrences of TEAE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of TEAE within a PT will be counted only once in that PT. Percentages will be based on the number of subjects in the safety analysis set.
- Summary tables for (5) and (6) A subject with multiple occurrences of TEAE within a SOC or a PT will be counted only once for the TEAE with the maximum intensity. Percentages will be based on the number of subjects in the safety analysis set.
- Property of Takedai. For none Summary table for (9) A subject with a TEAE that occurs in more than one interval is counted in all the intervals that the TEAE occurs. For each time interval, a subject with multiple occurrences of TEAE within a SOC or a PT will be counted only once in that SOC or PT. When calculating percentages for each time interval, the number of subjects at risk (i.e., subjects who either have an exposure or have an occurrence of TEAE, during or after the corresponding time interval) will be used as the denominator. The number of

,ble Terms of Use subjects whose onset of any one of the TEAEs is within the time interval will be used as the numerator.

#### 6.8.1.3 Displays of Pretreatment Events

Analysis Set: All Subjects Who Signed the Informed Consent Form

Analysis Endpoint(s): PTE

The following summaries will be provided using frequency Analytical Method(s):

distribution.

PTEs will be coded using the MedDRA and will be summarized using SOC and PT. SOC will be sorted alphabetically and PT will be sorted in decreasing frequency.

(1) Pretreatment Events by System Organ Class and Preferred Term

(2) Serious Pretreatment Events by System Organ Class and Preferred Term

The frequency distribution will be provided according to the rules below.

Number of subjects

A subject with multiple occurrences of PTE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of PTE within a PT will be counted only once in that PT.

#### 6.8.2 Clinical Laboratory Evaluations

6.8.2.1 Laboratory Tests other than Urinalysis

Analysis Set: Safety Analysis Set

Analysis Endpoint(s): See Section 9.3.6.

Visit: Using the visits (Baseline to Week 26) of the visit window defined in

Section 9.2.2.

Analytical Method(s): For each endpoint, summaries (1) to (3) will be provided.

(1) Summary of Laboratory Test Results and Change from Baseline

by Visit

Descriptive statistics for observed values and changes from baseline (each post-baseline visit - Baseline) will be provided for

each visit.

(2) Case Plots

Plots over time for each subject will be presented.

(3) Summary of Shifts of Laboratory Test Results Shift tables showing the number of subjects in each category at baseline and each post-baseline visit will be provided. For each laboratory test, the laboratory values will be classified as "Low", "Normal" or "High" relative to the normal reference range provided by the central laboratory. The shift tables will be based on these classifications.

#### 6.8.2.2 Urinalysis

Safety Analysis Set Analysis Set: Analysis Endpoint(s): See Section 9.3.6.

Using the visits (Baseline to Week 26) of the visit window defined in Visit:

Section 9.2.2.

For pH and specific gravity, summaries (1), (2) and (4) will be Analytical Method(s): provided.

> For each endpoint other than pH and specific gravity, summaries (3) and (4) will be provided.

- (1) Summary of Urine Laboratory Test Results and Change from baseline (each post-baseline visit - Baseline) will be provided for
- Shift tables showing the number of subjects in each category at
- A change in the control of the contr Shift tables showing the number of subjects in each category at classified as "Low", "Normal" or "High" relative to the normal

#### 6.8.3 Vital Signs, Weight and Height

Analysis Set: Safety Analysis Set

Systolic Blood Pressure Diastolic Blood Pressure Analysis Endpoint(s):

> Heart Rate **Body Temperature**

Weight Height

BMI Respiration Rate

Visit: Using the visits (Baseline to Week 26) of the visit window defined in

Section 9.2.2.

For each endpoint, summaries (1) and (2) will be provided. Analytical Method(s):

(1) Summary of Vital Signs, Weight and Height, and Change from

Baseline by Visit

Descriptive statistics for observed values and changes from baseline (each post-baseline visit - Baseline) will be provided for

each visit.

(2) Case Plots

Plots over time for each subject will be presented.

#### 6.8.4 **ECGs**

Safety Analysis Set Analysis Set:

Heart Rate Analysis Endpoint(s):

> RR Interval PR Interval **QRS** Interval **OT** Interval

**OTcF** Interval

Interpretation [Within Normal Limits, Abnormal but not

Clinically Significant, Abnormal and

Clinically Significant]

Analytical Method(s): Using the visits (Baseline to Week 26) of the visit window defined in

Section 9.2.2.

For each endpoint other than 12-lead ECG interpretations, summaries

(1) and (2) will be provided.

For ECG interpretation, summary (3) will be provided.

(1) Summary of ECG Parameters and Change from Baseline by Visit Descriptive statistics for observed values and changes from

baseline (each post-baseline visit - Baseline) will be provided for each visit.

(2) Case Plots
Plots over time for each subject will be presented.

(3) Summary of Shift of ECG Interpretation
Shift table showing the number of subjects in each category at baseline and each post-baseline visit will be provided.

## 6.8.5 Displays of Treatment-Emergent Adverse Events (Japanese)

Analysis Set: Safety Analysis Set

Analysis Endpoint(s): TEAE

Analytical Method(s): TEAEs will be summarized in the same way as in Section 6.8.1.2. All

summaries will be presented in Japanese.

### 6.9 Pharmacokinetic, Pharmacodynamic, and Biomarker Analyses

#### 6.9.1 Pharmacokinetic Analysis

6.9.1.1 Plasma Concentrations

Analysis Set: Safety Analysis Set

Analysis Endpoint(s): Plasma concentrations of TAK-625

Visit: Using the visits of the visit window defined in Section 9.2.2.2

Analytical Method(s): The following summaries will be provided.

(1) Summary of Plasma Concentrations by Visit Descriptive statistics will be provided by visit by dose level categories administered just before sample collection.

## 6.10 Other Analyses

#### 6.10.1 Analyses for Overall Supplemental Cohort

Cohort: Overall Supplemental Cohort

Analytical Method(s): The same analyses in section  $6.3 \sim 6.9$  will be performed for overall

supplemental cohort.

#### 6.10.2 Analyses for All Cohorts Combined

Cohort: All Cohorts Combined

- TEFERENCES

  [1] World Health Organization (WHO) growth charts "A SAS Program for the WHO Growth Charts (ages 0 to < 2 years)"

  https://www.cdc.gov/nccdphp/dnpao/growthcharts/resources/sec = 1

  [2] Centers for Disease Control (CDC)

  Growth CL
- Growth Charts (ages 0 to < 20 years)" https://www.cdc.gov/nccdphp/dnpao/growthcharts/resources/sas.htm

#### CHANGES TO PROTOCOL PLANNED ANALYSES 8.0

There was no change to the protocol planned analyses.

#### 9.0 **APPENDIX**

#### Changes From the Previous Version of the SAP 9.1

From the SAP version 1.0, the major updates except minor updates like error correction were following parts.

Section

Before the change

Not applicable.

After the change



Reason for the change

Some exploratory endpoints were added when protocol had been amended.

Section 6.0 STATISTICAL ANALYSIS

Before the change

Not applicable.

After the change

ot to the applicable Ter Statistical analyses will be performed using all subjects' data up to Week 26 (i.e., up to Day 197) after the data are locked. PK analysis will be performed using all subjects' data up to Week 10 after the data are locked.

Reason for the change

To make the target range of the Interim analysis clear.

Section 6.1 General Considerations

Before the change

- Descriptive statistics: Number of subjects, mean, standard deviation, standard error, maximum, minimum, and quartiles (Q1, median, and Q3).
- Duration of exposure to study drug (days): Date of last dose of study drug date of first dose of study drug + 1.
- Duration of study after baseline (days): Date of last visit/contact date of first dose of study drug + 1.
- **Time to liver-associated events:** PEBD surgery, listing for liver transplantation, liver decompensation [hepatic encephalopathy, variceal bleeding, ascites, and spontaneous bacterial per.
  After the change bacterial peritonitis] events, hepatocellular carcinoma (HCC), death.

- Descriptive statistics for endpoints other than PK: Number of subjects, mean, standard deviation, standard error, maximum, minimum, and quartiles (Q1, median, and Q3).
- **Descriptive statistics for PK**: Number of subjects, mean, standard deviation, maximum, median, minimum, coefficient of variation, and geometric mean.

- **Duration of exposure to study drug (days)**: {Date of last dose of study drug or Week 26 visit (i.e. the latest visit by Day 197) which comes faster date of first dose of study drug} + 1.
- **Duration of study after baseline (days)**: {Date of last visit/contact or Week 26 visit (i.e. the latest visit by Day 197) which comes faster date of first dose of study drug} + 1.

••

- Dose Level (μg/kg): Strength of study drug taken (mg) / (last available body weight (kg) prior to or on the day of study drug taken) \* 1000.
- Dose Level Categories for PK ( $\mu$ g/kg): Categorize by following below calculation rule. If Min <= dose level < 225  $\mu$ g/kg, then dose level category = 150  $\mu$ g/kg; if 225  $\mu$ g/kg <= dose level < 375  $\mu$ g/kg, then dose level > category = 300  $\mu$ g/kg; if 375  $\mu$ g/kg <= dose level < 525  $\mu$ g/kg, then dose level category = 450  $\mu$ g/kg; if 525  $\mu$ g/kg <= dose level <= Max, then dose level category = 600  $\mu$ g/kg.
- Total Drug Exposure (μg/kg): Sum of {number of study drugs taken \* dose level received (μg/kg)}.
- Average Daily Dose (μg/kg/day): Total Drug Exposure (μg/kg) / Duration of exposure to study drug (days).

. . .

• **Time to liver-associated events**: PEBD surgery, listing for liver transplantation, liver decompensation [hepatic encephalopathy, variceal bleeding, ascites, and spontaneous bacterial peritonitis] events, hepatocellular carcinoma (HCC), death, and other.

. . .

- Corrected Sodium (mEq/L): sodium (mEq/L) + (0.002 \* Triglycerides (mg/dL)).
- FIB-4: (Age (years) \* AST (U/L)) / (platelet count  $(10^9/L)$  \* sqrt(ALT(U/L)))
  - Age (years) is years at sample collection visit.
- APRI: 100 \* (AST (U/L) / AST ULN(U/L)) / (platelet count (10^9/L))
  - > <u>ULN is upper limit normal</u>
- Significant Protocol Deviation: Deviation defined in the PDMP as "Important PD" whose Severity Classifications is "major" or "critical".
- <u>Time since original diagnosis of PFIC (months)</u>: (date of first dose date of original diagnosis of PFIC + 1) / 30.4375.

Reason for the change

Some calculation rules and definitions were added and updated.

Before the change

Not applicable.

After the change

When reporting derived values or parameters, following presenting rules will be applied.

- For sBA, ItchRO: For rules on rounding and decimal presentation of these statistics, along with the rules for presenting certain derived values see below.
  - For measures of median and mean, use 3 decimal places.
  - For measures of standard deviation, standard error of the mean and CL use 4 decimal places.
  - For measures of minimum and maximum values as well as observed value (for Listing), use 2 decimal places.
  - >=5 is rounded up away from zero, whereas <5 is rounded down toward zero, to account for rounding of negative numbers.
  - For p-values use 3 decimal places.
  - > Presentation of p-values display p-values that would round to 0.000 as <0.001.
- Other than sBA, and ItchRO: For rules on rounding and decimal presentation of these statistics, along with the rules for presenting certain derived values see below.
  - For measures of median and mean, use 1 decimal place beyond those used for the measurement.
  - For measures of standard deviation, standard error of the mean and CI, use 2 decimal places beyond those used for the measurement.
  - For measures of minimum and maximum values, use the same number of decimal places as those used for the measurement.
  - >=5 is rounded up away from zero, whereas <5 is rounded down toward zero, to account for rounding of negative numbers.
  - For p-values use 3 decimal places.
  - Presentation of p-values display p-values that would round to 0.000 as <0.001.
  - BMI should be rounded to 1 decimal place for reporting.
  - Derived questionnaire scores, and other similar efficacy parameters recorded as integers, should be rounded to 1 decimal place for reporting.
  - Averaged lab results (e.g. Diastolic/Systolic Blood Pressure and Pulse [when taken in triplicate]) should be rounded to 1 decimal place for reporting.

Reason for the change

Presenting rules in TLF were added.

Section 6.3.2 Screen Failures

Before the change

Analysis Endpoint(s): Age (months)

After the change

Not applicable.

Reason for the change

No infant subjects who failed screening.

Section 6.3.5 Disposition of Subjects

Before the change

to the applicable Terrins of Use Analysis Endpoint(s): Study Drug Administration Status, [Eligible but Not Treated]

Reason for Not Being Treated, [AE, Screen Failure (Did not meet inclusion criteria or did meet exclusion criteria), Protocol Deviation, Lost to Follow-up, Pregnancy, Withdrawal by Subject, Study Terminated by Sponsor, Other]

Study Drug Completion Status, [Completed Study Drug, Prematurely Discontinued Study Drug]

Completion Status of All Planned Study Visits, Completed Study, Prematurely Discontinued Study]

Analytical Method(s): Frequency distributions will be provided. When calculating percentages for the reasons for not being treated, the total number of subjects not treated by the study drug will be used as the denominator. When calculating percentages for the reasons for discontinuation, the total number of subjects who prematurely discontinued will be used as the denominator.

After the change

Analysis Endpoint(s):

Study Drug Completion Status, [Ongoing, Completed Study Drug, Prematurely Discontinued Study Drug

Completion Status of All Planned Study Visits, [Ongoing, Completed Study, Prematurely Discontinued Study]

Analytical Method(s): Frequency distributions will be provided. When calculating percentages for the reasons for discontinuation, the total number of subjects who prematurely discontinued will be used as the denominator.

Reason for the change

These analysis endpoints were not appropriate for ITT population. The category of "Ongoing" was added because this SAP is for Interim analysis.

Section 6.3.6.1 Significant Protocol Deviations

Before the change

Analysis Endpoint(s): Significant Protocol Deviations, [AE, Screen Failure (Did not meet inclusion criteria or did meet exclusion criteria), Protocol Deviation, Lost to Follow-up, Pregnancy, Withdrawal by Subject, Study Terminated by Sponsor, Other]

After the change

Analysis Endpoint(s): Significant Protocol Deviations, [Informed Consent and Process, Inclusion Criteria, Exclusion Criteria, Concomitant Medication, Laboratory Assessment, Study Procedures (not safety and efficacy related), Safety, Visit Schedule, IP conditions, IP preparation, IP administration, Subject IP Compliance, Efficacy, Subject Discontinuation, Administrative, Patient Reported Outcomes, PK/PD, Other Criteria]

Reason for the change

Change it from CRF category to CTMS category.

Section 6.4.1 Demographic and Baseline Characteristics

Before the change

Analysis Endpoint(s): Age (years), [Min<= - < 9, 9<= - <=18, 18< - <=Max]

After the change

Analysis Endpoint(s): Age (years), [Min<= - < 9, 9<= - <=18, 18< - <=Max]

 $[Min \le - <7, 7 \le - \le Max]$ 

Reason for the change

Added CTD analysis category.

Section 6.6 Extent of Exposure and Compliance

Before the change

Analysis Endpoint(s): Not applicable.

Analytical Method(s): (1) Study Drug Exposure and Compliance

After the change

Analysis Endpoint(s): <u>Total Drug Exposure (μg/kg)</u>, <u>Average Daily Dose (μg/kg/day)</u>

Analytical Method(s): (1) Study Drug Exposure, Compliance, Total Drug Exposure and

Average Daily Dose

Reason for the change

Added additional endpoints.

Section

Before the change

Analysis Endpoint(s):

After the change

Analysis Endpoint(s):

Reason for the change

Added new exploratory endpoints when protocol had been amended.

Section 6.7.3.3 Responder Analysis
Before the change

Not applicable.

After the change

Analysis Set:, ITT



Reason for the change

Added new exploratory endpoints when protocol had been amended.

Section 6.7.4 Subgroup Analysis

Before the change

Subgroup(s): Age, [Min<= - < 9, 9<= - <=18, 18< - <=Max]

After the change

Subgroup(s): Age, [Min $\leq$  -  $\leq$  - < -

Reason for the change

To be consistent with CTD analysis.

Section 6.9.1.1 Plasma Concentrations

Before the change

Analytical Method(s): The following summaries will be provided.

(1) Summary of Plasma Concentrations by Visit Descriptive statistics will be provided.

After the change

Analytical Method(s): The following summaries will be provided.

(1) Summary of Plasma Concentrations by Visit Descriptive statistics will be provided by visit by dose level categories administered just before sample collection.

Reason for the change

To incorporate new Clinical pharmacology insight.

Section 9.2.1 Definition of Study Days

Before the change

The following definitions and calculation formulas will be used.

- Study Day: The day before the first dose of the study drug will be defined as Study Day -1 and the day of the first dose will be defined as Study Day 1. If the date of the observation is on the same date or after the day of the first dose, Study Day will be calculated relative to Study Day 1. Otherwise, Study Day will be calculated relative to Study Day -1.
- Follow-up Day: The day after the last dose of the study drug will be defined as Follow-up Day 1. Follow-up Day will be calculated relative to Day 1.

After the change

The following definitions and calculation formulas will be used.

- Study Day: The day before the first dose of the study drug will be defined as Study Day -1 and the day of the first dose will be defined as Study Day 1. If the date of the observation is on the same date or after the day of the first dose, Study Day will be calculated relative to Study Day 1. Otherwise, Study Day will be calculated relative to Study Day -1.
- Follow-up Day: The day after the last dose of the study drug will be defined as Follow-up Day 1.

Reason for the change

Error correction.

Section 9.2.2.1 Endpoints other than ItchRO Scores and PK Samples

Before the change

For each visit, observation obtained in the corresponding time interval will be used. If more than one observation lies within the same visit window, the observation with the closest Study Day to the scheduled Study Day will be used. If there are two observations equidistant to the scheduled Study Day, the later observation will be used.

After the change

For each visit, observation obtained in the corresponding time interval will be used. If more than one observation lies within the same visit window, the observation with the closest Study Day to the scheduled Study Day will be used. If there are two observations equidistant to the scheduled Study Day, the later observation will be used. For laboratory test data, if there are two observations of both central laboratory sample and local sample on the same date, central

laboratory sample data will be used. Values less than or equal to the lower limit of quantification applicable Terms of will be treated as one-half of the lower limit value when calculating the descriptive statistics. Values greater than or equal to the upper limit of quantification will be treated as the upper limit value when calculating the descriptive statistics.

Reason for the change

Added handling rule for the lower limit of quantification value.

#### Section 9.2.2.2 PK Samples

#### Before the change

Study Time (hour) is defined as the difference from the PK sampling time at the visit date to the time of study drug taken at the visit date (rounded to 1 decimal place(s)).

For each visit, observation obtained in the corresponding time interval will be used. If more than one observation lies within the same visit window, the observation with the closest Study Time to the scheduled Study Time will be used. If there are two observations equidistant to the scheduled Study Time, the earlier observation will be used.

Visit Window of PK Table 9.8

| Visit | Da | ed Study<br>ay<br>ys) | Time Interval (days) Study Day | Scheduled Study<br>Time | Study<br>Time<br>(hours) |
|---|---|---|---|---|---|
| Pre-dose at Week 10 | Study<br>Day: | 71 | 71 | Study<br>Time 0<br>(hour): | -5.0 ~<br>0.0 |
| 2.5 Hours after<br>Morning Dose at<br>Week 10 | Study<br>Day: | 71 | 71 | Study<br>Time 2.5<br>(hour): | 1.5 ~ 3.5 |
| Pre-dose at Week 14 ~ 26 | <u>Study</u><br><u>Day:</u> | <u>99</u> | <u>99 – 183</u> | Study<br>Time 0<br>(hour): | <u>-5.0 ~</u><br><u>0.0</u> |
| 0.5 Hours after Morning Dose at Week 14 ~ 26 | <u>Study</u><br><u>Day:</u> | 99 | <u>99 – 183</u> | <u>Study</u><br><u>Time</u> <u>0.5</u><br>(hour): | <u>0.0 ~ 1.0</u> |

After the change

Study Time (hour) is defined as the difference from the PK sampling time at the visit date to the time of study drug taken at the visit date (rounded to 1 decimal place(s)).

For each visit, observation obtained in the corresponding time interval will be used. If more than one observation lies within the same visit window, the observation with the closest Study Time to the scheduled Study Time will be used. If there are two observations equidistant to the scheduled Study Time, the earlier observation will be used. Values less than the lower limit of quantification will be treated as zero when calculating the descriptive statistics.

| Visit | D | ed Study<br>ay<br>ys) | Time Interval<br>(days)<br>Study Day | Scheduled Study Time | Study<br>Time<br>(hours) |
|---|---|---|---|---|---|
| Pre-dose at Week 10 | Study<br>Day: | 71 | <u>57 - 85</u> | Study Time 0 (hour): | -5.0 ~<br>0.0 |
| 2.5 Hours after<br>Morning Dose at<br>Week 10 | Study<br>Day: | 71 | 57 - 85 and | Study<br>Time 2.5<br>(hour): | 1.5 ~ 3.5 |

Reason for the change

Added handling rule for the lower limit of quantification value. For Visit window, some Visits were removed because it's possible that samples at these visits not to be collected at Interim analysis. For Time interval, previous one was too narrow and inappropriate.

Section 9.2.3 Partial Date Conventions

Before the change

Not applicable.

After the change

### 9.2.3 Partial Date Conventions

For Medication History and Concomitant Medication, if their stop date is partially/completely missing, following handling rules will be applied.

if (CMCAT="MEDICATION HISTORY") then "(1) Prior Medication";

else if (CMENRTPT="ONGOING") then "(3) Concomitant Medication":

else if

(. < medication end year < TAK-625 start year) or

medication end year = TAK-625 start year and . < medication end month < TAK-625 start month) or medication end year = TAK-625 start year and medication end month = TAK-625 start month and . < medication end date < TAK-625 start date ) then "(2) Concomitant Medication" ect to the application else "(3) Concomitant Medication";

Reason for the change

To make it clear how to handle partial date.

Section 9.3.2 Average ItchRO Scores

Before the change

Both the morning and evening ItchRO reports have a minimum score of 0 and a maximum score of 4, with 4 representing more severe (Item 1) or more frequent (Item 3) itching. After the derivation described in section 9.2.2.3, the following endpoints will be derived the same procedures as section 9.3.1.

- Change in the average evening ItchRO (Obs/Pt) severity score between baseline and average of Week 15 through Week 26.
- Change in the average ItchRO (Obs/Pt) severity (based on daily maximum of morning and evening severity scores)
- Change in the average morning ItchRO (Obs/Pt) frequency score between baseline and average of Week 15 through Week 26.
- Change in the average evening ItchRO (Obs/Pt) frequency score between baseline and average of Week 15 through Week 26.

After the change

For ItchRO scores, both the morning and evening ItchRO reports have a minimum score of 0 and a maximum score of 4, with 4 representing more severe (Item 1) or more frequent (Item 3) itching. After the derivation described in section 9.2.2.3, the following endpoints will be derived the same procedures as section 9.3.1.

- Change in the average evening ItchRO (Obs/Pt) severity score between baseline and average of Week 15 through Week 26.
- Change in the average ItchRO (Obs/Pt) severity and frequency (based on daily maximum of morning and evening severity scores) between baseline and average of Week 15 through Week 26.
- Change in the average morning ItchRO (Obs/Pt) frequency score between baseline and average of Week 15 through Week 26.
- Change in the average evening ItchRO (Obs/Pt) frequency score between baseline and average of Week 15 through Week 26.

Reason for the change

Added new exploratory endpoints when protocol had been amended.

Section 9.3.3 Responder Endpoints

Before the change

• **Subjects who experience an sBA control**: subjects with a reduction to <102 μMol/L, or a reduction of >75%, or normalization) from baseline through Week 26

After the change

• Subjects who experience an sBA control: subjects with a reduction to <102 μMol/L, or a reduction of >75%, or normalization) from baseline through Week 26





Reason for the change

commercial use only and sul Added new exploratory endpoints when protocol had been amended.

Section 9.3.6 Lists of Laboratory Tests

Before the change

Not applicable.

After the change

Total sBA (enzymatic assay)

Reason for the change

Error correction.

#### **Data Handling Conventions** 9.2

#### **Definition of Study Days** 9.2.1

The following definitions and calculation formulas will be used.

- Study Day: The day before the first dose of the study drug will be defined as Study Day -1 and the day of the first dose will be defined as Study Day 1. If the date of the observation is on the same date or after the day of the first dose, Study Day will be calculated relative to Study Day 1. Otherwise, Study Day will be calculated relative to Study Day -1.
- Follow-up Day: The day after the last dose of the study drug will be defined as Follow-up Day 1.

#### 9.2.2 Definition of Study Visit Windows

When calculating Study Day relative to a reference date (i.e., date of first dose of study drug [Day 1]), if the date of the observation is on the same date or after the reference date, it will be calculated as: date of observation - reference date + 1; otherwise, it will be calculated as: date of observation - reference date. Hence, reference day is always Day 1 and there is no Day 0.

When calculating Follow-up Day relative to a reference date (i.e., date of last dose of study drug [Follow-up Day 0]), it will be calculated as: date of observation - reference date. Hence, reference day is always Follow-up Day 0.

All evaluable data (i.e., non-missing data) will be handled according to the following rules.

### 9.2.2.1 Endpoints other than ItchRO Scores and PK Samples

For each visit, observation obtained in the corresponding time interval will be used. If more than one observation lies within the same visit window, the observation with the closest Study Day to the scheduled Study Day will be used. If there are two observations equidistant to the scheduled Study Day, the later observation will be used. For laboratory test data, if there are two observations of both central laboratory sample and local sample on the same date, central laboratory sample data will be used. Values less than or equal to the lower limit of quantification will be treated as one-half of the lower limit value when calculating the descriptive statistics. Values greater than or equal to the upper limit of quantification will be treated as the upper limit value when calculating the descriptive statistics.

Table 9.1 Visit Window of sBA, BA subspecies, C4, Serum Storage Sample

| 77:-:4 | Scheduled Study Day | Time Interval (days) | |
|---|---|---|---|
| Visit | (days) | Study Day | Follow-up Day |
| Baseline (Week 0) | Study Day: 1 | -42 - 1 | |
| Week 2 | Study Day: 15 | 2 - 29 | < 15 |
| Week 6 | Study Day: 43 | 30 - 57 | < 15 |
| Week 10 | Study Day: 71 | 58 - 85 | < 15 |
| Week 14 | Study Day: 99 | 86 - 113 | < 15 |
| Week 18 | Study Day: 127 | 114 - 141 | < 15 |
| Week 22 | Study Day: 155 | 142 - 169 | < 15 |
| Week 26 | Study Day: 183 | 170 - 197 | < 15 |

Table 9.2 <u>Visit Window of Vital Signs, Weight</u> and Height,

| 77:-:4 | Scheduled Study Day | Time Inter | val (days) |
|-------------------|---------------------|------------|---------------|
| Visit | (days) | Study Day | Follow-up Day |
| Baseline (Week 0) | Study Day: 1 | -42 - 1 | Ne |
| Week 2 | Study Day: 15 | 2 - 22 | (CO < 15 |
| Week 4 | Study Day: 29 | 23 - 36 | < 15 |
| Week 6 | Study Day: 43 | 37 - 57 | < 15 |
| Week 10 | Study Day: 71 | 58 - 85 | < 15 |
| Week 14 | Study Day: 99 | 86 - 113 | < 15 |
| Week 18 | Study Day: 127 | 114 - 141 | < 15 |
| Week 22 | Study Day: 155 | 142 - 169 | < 15 |
| Week 26 | Study Day: 183 | 170 - 197 | < 15 |

Table 9.3 Urinalysis, Cholestasis Biomarkers (FGF19)

| 77 | Scheduled Study Day | Time Interval (days) | |
|---|---|---|---|
| Visit | (days) | Study Day | Follow-up Day |
| Baseline (Week 0) | Study Day: 1 | -42 - 1 | |
| Week 6 | Study Day: 43 | 2 - 57 | < 15 |
| Week 10 | Study Day: 71 | 58 - 99 | < 15 |
| Week 18 | Study Day: 127 | 100 - 155 | < 15 |
| Week 26 | Study Day: 183 | 156 – 197 | < 15 |

Table 9.4 Lipid Panel, Lipid Soluble Vitamins

| ##1 14 | Scheduled Study Day | Time Inter | val (days) |
|-------------------|---------------------|-----------------|---------------|
| Visit | (days) | Study Day | Follow-up Day |
| Baseline (Week 0) | Study Day: 1 | <b>-</b> 42 – 1 | |

Lipid Panel, Lipid Soluble Vitamins Table 9.4

| T7"'4 | Scheduled Study Day | Time Interval (days) | |
|---------|---------------------|----------------------|---------------|
| Visit | (days) | Study Day | Follow-up Day |
| Week 6 | Study Day: 43 | 2 – 57 | < 15 |
| Week 10 | Study Day: 71 | 58 – 85 | 15 |
| Week 14 | Study Day: 99 | 86 – 113 | < 15 |
| Week 18 | Study Day: 127 | 114 – 141 🗷 | < 15 |
| Week 22 | Study Day: 155 | 142 - 169 | < 15 |
| Week 26 | Study Day: 183 | 170 – 197 | < 15 |

Table 9.5

| | 1 | 157 | |
|------------------------|------------------------|------------|---------------|
| Table 9.5 CBC, Coagula | ation, Chemistry Panel | sulos | |
| X7114 | Scheduled Study Day | Time Inter | val (days) |
| Visit | (days) | Study Day | Follow-up Day |
| Baseline (Week 0) | Study Day: 1 | -42 - 1 | |
| Week 2 | Study Day: 15 | 2 - 29 | < 15 |
| Week 6 | Study Day: 43 | 30 - 57 | < 15 |
| Week 10 | Study Day: 71 | 58 - 85 | < 15 |
| Week 14 | Study Day: 99 | 86 - 113 | < 15 |
| Week 18 | Study Day: 127 | 114 - 141 | < 15 |
| Week 22 | Study Day: 155 | 142 - 169 | < 15 |
| Week 26 | Study Day: 183 | 170 - 197 | < 15 |

Visit Window of ECGs, AFP

| Visit | | Scheduled Study Day | Time Interval (days) | |
|---|---|---|---|---|
| | | (days) | Study Day | Follow-up Day |
| Baseline (Week | 0) | Study Day: 1 | -42 - 1 | |

Table 9.6 Visit Window of ECGs, AFP

| X7"'4 | Scheduled Study Day | Time Inter | val (days) |
|---------|---------------------|------------|---------------|
| Visit | (days) | Study Day | Follow-up Day |
| Week 10 | Study Day: 71 | 2 - 127 | < 15 |
| Week 26 | Study Day: 183 | 128 - 197 | ₹ 15 |



## 9.2.2.2 PK Samples

Study Time (hour) is defined as the difference from the PK sampling time at the visit date to the time of study drug taken at the visit date (rounded to 1 decimal place(s)).

For each visit, observation obtained in the corresponding time interval will be used. If more than one observation lies within the same visit window, the observation with the closest Study Time to the scheduled Study Time will be used. If there are two observations equidistant to the scheduled Study Time, the earlier observation will be used. Values less than the lower limit of quantification will be treated as zero when calculating the descriptive statistics.

Table 9.8 Visit Window of PK

| Visit | D | ed Study<br>ay<br>ays) | Time Interval<br>(days)<br>Study Day | Scheduled Study<br>Time | Study<br>Time<br>(hours) |
|---|---|---|---|---|---|
| Pre-dose at Week 10 | Study<br>Day: | 71 | 57 - 85 | Study Time 0 (hour): | -5.0 ~<br>0.0 |
| 2.5 Hours after<br>Morning Dose at<br>Week 10 | Study<br>Day: | 71 | 57 - 85 | Study<br>Time 2.5<br>(hour): | 1.5 ~ 3.5 |

### 9.2.2.3 Average ItchRO Scores

For each visit other than Week 6, average ItchRO score is defined as the average of the scores (morning, evening, or daily maximum of morning and evening) over the visit consisting of the 28 days on or before the scheduled Study Day (i.e., the sum of the scores divided by the number of non-missing scores). The answer "I don't know" will be treated as missing.

For Week 6, average ItchRO score is defined as the average of the scores (morning, evening, or daily maximum of morning and evening) over the visit consisting of the 41 days on or before the scheduled Study Day (i.e., the sum of the scores divided by the number of non-missing scores). The answer "I don't know" will be treated as missing.

In the event that a subject caregiver failed to complete the morning/evening report, the morning/evening score for that day will be treated as missing data. If 25% or more ItchRO scores for the post-baseline visit are missing, the average ItchRO score at that visit will be treated as missing. The restriction is not set for baseline average ItchRO scores.

158

| 77' '/ | Scheduled Study Day | Time Interval (days) | |
|---|---|---|---|
| Visit | (days) | Study Day | Follow-up Day |
| Baseline (Week 0) | Study Day: -1 | -281 | <0, |
| Week 6 | Study Day: 42 | 2 - 42 | ≥ 15 |
| Week 10 | Study Day: 70 | 43 - 70 | < 15 |
| Week 14 | Study Day: 98 | 71 - 98 | < 15 |
| Week 18 | Study Day: 126 | 99 - 126 | < 15 |
| Week 22 | Study Day: 154 | 127 - 154 | < 15 |
| Week 26 | Study Day: 182 | 155 - 182 | < 15 |

Table 9.9 Visit Window of Average ItchRO Score

#### 9.2.3 Partial Date Conventions

For Medication History and Concomitant Medication, if their stop date is partially/completely missing, following handling rules will be applied.

#### 9.3 Derivation of Endpoints

#### 9.3.1 Primary Efficacy Endpoints

Both the morning and evening ItchRO reports have a minimum score of 0 and a maximum score of 4, with 4 representing more severe (Item 1) itching. The derivation method for the primary efficacy endpoint will be described below.

After the derivation described in section 9.2.2.3, each subject will have a baseline (Week 0) average morning ItchRO (Obs) severity score, and have post-baseline average morning ItchRO (Obs) severity scores at Weeks 18, Week 22, and Week 26. For each subject, change in the average morning ItchRO (Obs) severity score between baseline and post-baseline visit can be calculated at Weeks 18, Week 22, and Week 26. Hence, the primary efficacy endpoint for each subject can be calculated as an average of the changes in the average morning ItchRO (Obs) severity score from Week 15 through Week 26 (i.e., the sum of the average morning ItchRO (Obs) severity scores divided by the number of non-missing morning severity scores).

### 9.3.2 Average ItchRO Scores

For ItchRO scores, both the morning and evening ItchRO reports have a minimum score of 0 and a maximum score of 4, with 4 representing more severe (Item 1) or more frequent (Item 3) itching. After the derivation described in section 9.2.2.3, the following endpoints will be derived the same procedures as section 9.3.1.



- Change in the average evening ItchRO (Obs/Pt) severity score between baseline and average of Week 15 through Week 26.
- Change in the average ItchRO (Obs/Pt) severity and frequency (based on daily maximum of morning and evening severity scores) between baseline and average of Week 15 through Week 26.
- Change in the average morning ItchRO (Obs/Pt) frequency score between baseline and average of Week 15 through Week 26.
- Change in the average evening ItchRO (Obs/Pt) frequency score between baseline and average of Week 15 through Week 26.

## 9.3.3 Responder Endpoints

• Subjects who experience an sBA control: subjects with a reduction to  $<102 \mu Mol/L$ , or a reduction of >75%, or normalization) from baseline through Week 26





#### 9.3.5

Z-scores of weight, height and BMI are based on a subject's gender and age at each scheduled visit. For subjects less than 24 months of age, the World Health Organization (WHO) growth charts are recommended by the Centers for Disease Control (CDC) and will be used to derive zscores. For subjects at least 24 months of age, the CDC growth charts will be used to derive zscores.

age at which he age at baseline. Age at which height and weight were measured should be used for calculating z-scores, not using

### 9.3.6 Lists of Laboratory Tests

| H(CDC'41- | Characteristics | T'.'IDI | TI. ''. |
|---|---|---|---|
| Hematology (CBC with | <u>Chemistry</u> | <u>Lipid Panel</u> | <u>Urinalysis</u> |
| <u>Differential</u> ) | Albumin | Total cholesterol | рН |
| Hematocrit | ALP | LDL-C (direct) | Specific gravity |
| Hemoglobin | Amylase | HDL-C | Protein |
| MCV, MCH, MCHC | ALT (SGPT) | TG | Specific gravity Protein Glucose Ketones |
| Red blood cells | AST (SGOT) | | Ketones |
| Platelets | Bicarbonate | <b>Cholestasis Biomarkers</b> | Bilirubin C |
| White blood cells | Bilirubin, direct | sBA (LC-MS) | Occult blood and cells |
| WBC Differential (% and | (conjugated) | sBA subspecies | Nitrite |
| absolute) | TSB | 7alpha-hydroxy-4- | Urobilinogen |
| Neutrophils | BUN | cholesten-3-one (C4) | Leukocyte esterase |
| Eosinophils | Calcium | FGF-19 | Microscopic examination |
| Basophils | Chloride | Autotaxin | Oxalate |
| Lymphocytes | Creatinine | .0) | Urinary creatinine |
| Monocytes | GGT | Lipid Soluble | , |
| | Glucose | <u>Vitamins</u> | |
| <u>Coagulation</u> | Lipase | 25-hydroxy vitamin D | |
| aPTT (sec) | Phosphate | Retinol | |
| INR | Potassium | RBP | |
| PT (sec) | Sodium | Alpha-tocopherol | |
| | Corrected Sodium | Estimated Total Lipids | |
| | Total protein | Ratio of Alpha-tocopherol | |
| | Total sBA (enzymatic assay) | to Estimated Total Lipids | |
| | Uric Acid | | |
| | Measured serum Osmolality | | |

## 9.3.7 Table for AECI

The categories of AECI will follow ones in CRF.

# 9.3.8 Significance Level and Confidence Coefficient

• Significance level: 5% (two-sided)

Confidence coefficient: 95% (two-sided)

## 9.4 Analysis Software

SAS (version 9.4)